CLINICAL TRIAL: NCT02831764
Title: A Phase III, Randomised, Double-blind, Multicentre, Parallel-group, Non-inferiority Study Evaluating the Efficacy, Safety, and Tolerability of Dolutegravir Plus Lamivudine Compared to Dolutegravir Plus Tenofovir/Emtricitabine in HIV-1-infected Treatment-naïve Adults
Brief Title: An Efficacy, Safety, and Tolerability Study Comparing Dolutegravir (DTG) Plus Lamivudine (3TC) With Dolutegravir Plus Tenofovir/Emtricitabine in Treatment naïve HIV Infected Participants (Gemini 2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205543; 2016-000459-28 (EudraCT Number)
Record Dates: First submitted 2016-07-08; First posted 2016-07-13 (Estimated); Results first posted 2019-04-22 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Infection, Human Immunodeficiency Virus; HIV Infections
Keywords: tolerability; HIV 1; efficacy; treatment naïve; two-drug regimen; safety; non inferiority
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome; HIV Infections | interventions — dolutegravir; Lamivudine; Tenofovir; Emtricitabine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DTG + 3TC (50 mg+300 mg (Experimental): Eligible participants will receive one 50 mg tablet of DTG plus one overencapsulated 300 mg 3TC tablet orally once daily upto 96 weeks; thereafter will receive DTG plus 3TC tablet upto Week 148 and will continue to receive this schedule until (i) DTG and 3TC are both locally approved for use as part of a dual regimen, and the single entities of DTG and 3TC are available to patients (e.g. through public health services), or (ii) the DTG/3TC FDC tablet, if required by local regulations, is available, , or (iii) the participant no longer derives clinical benefit, or (iv) the participant meets a protocol defined reason for discontinuation, or (v) development of the DTG plus 3TC dual regimen is terminated.
  Interventions: Drug: Dolutegravir (DTG); Drug: Lamivudine (3TC)
- DTG + TDF/FTC FDC (50 mg+300/200 mg) (Active Comparator): Eligible participants will receive one 50 mg tablet of DTG plus one overencapsulated TDF/ FTC FDC (300/200 mg) tablet orally once daily upto 96 weeks; thereafter will receive DTG plus TDF/FTC FDC tablets upto Week 148 (open-label randomised phase).
  Interventions: Drug: Dolutegravir (DTG); Drug: Tenofovir disoproxil fumarate/Emtricitabine (TDF/FTC FDC)

INTERVENTIONS:
Drug: Dolutegravir (DTG) — DTG is available as 50 mg white, round, biconvex, film coated tablet debossed on one side with 'SV 572' and on the other side with '50'. The tablets are packaged into high density polyethylene (HDPE) bottles with induction seals and child resistant closures. Each 45 ml bottle contains 30 tablets and a desiccant. DTG 50 mg tablet will be orally administered once daily with or without food upto 148 weeks.
Drug: Lamivudine (3TC) — Lamivudine is available as swedish orange, 'AA' sized elongated double blind HPMC capsules containing 300 mg lamivudine to visually match overencapsulated TDF/FTC FDC tablet. The capsules are packaged into HDPE bottles with induction seals and child resistant closures. Each 150 mL bottle contains 30 capsules and a desiccant. Overencapsulated 3TC 300 mg tablet will be orally administered once daily with or without food upto 96 weeks. From Week 96 to Week 148, lamivudine will be dispensed as 300 mg white, diamond shaped, scored, film coated tablets debossed with 'GX CJ7' on both sides, packed in over labelled HDPE bottles with child-resistant closures each containing 30 tablets.
  Arms: DTG + 3TC (50 mg+300 mg
Drug: Tenofovir disoproxil fumarate/Emtricitabine (TDF/FTC FDC) — Tenofovir disoproxil fumarate and Emtricitabine are available as swedish orange, 'AA' sized elongated double blind HPMC capsules containing 300 mg TDF and 200 mg FTC to visually match overencapsulated 3TC tablet. The capsules are packaged into HDPE bottles with induction seals and child resistant closures. Each 150 mL bottle contains 30 capsules and a desiccant. Overencapsulated tenofovir disoproxil fumarate/emtricitabine tablet will be orally administered once daily with or without food upto 96 weeks. From Week 96 to Week 148, tenofovir disoproxil fumarate/emtricitabine will be dispensed as 300/200 mg white, blue, capsule shaped, film coated tablets debossed with 'GILEAD' on one side and '701' on another side, packed in overlabelled HDPE bottles with polypropylene childresistant closures each containing 30 tablets and a desiccant.
  Arms: DTG + TDF/FTC FDC (50 mg+300/200 mg)

SUMMARY:
This study will compare safety, efficacy, and tolerability of a two drug regimen of dolutegravir (DTG) plus (+) lamivudine (3TC) administered once daily with DTG plus two nucleoside reverse transcriptase inhibitors (tenofovir disoproxil fumarate [TDF]/emtricitabine [FTC] fixed dose combination [FDC]) administered once daily in human immunodeficiency virus (HIV) 1 infected adult participants that have not previously received antiretroviral therapy. The study is designed to demonstrate the non inferior antiviral activity of DTG + 3TC regimen to that of DTG + TDF/FTC FDC and will characterise the long term antiviral activity, tolerability and safety of DTG plus 3TC through Week 148. Approximately, 700 participants will be randomised 1:1 to receive DTG + 3TC or DTG + TDF/FTC FDC. Participants will be stratified by screening HIV 1 ribonucleotide nucleic acid (RNA) levels and by screening CD4+ (cluster of differentiation 4) cell count.

ELIGIBILITY:
Inclusion Criteria:

* Must be an HIV 1 infected adult >=18 years of age (or older, if required by local regulations) at the time of signing the informed consent
* An eligible female participant should not be pregnant (as confirmed by a negative serum human chorionic gonadotrophin (hCG) test at Screening and negative urine test at Baseline), not lactating, and at least one of the following conditions applies

  * Non reproductive premenopausal women are those that have undergone documented tubal ligation or documented hysteroscopic tubal occlusion procedure with follow up confirmation of bilateral tubal occlusion or documented bilateral oophorectomy or hysterectomy
  * Non reproductive premenopausal women are those with 12 months of spontaneous amenorrhea and >=45 years of age
  * Women with reproductive potential agree to follow one of the protocol-defined methods for avoiding pregnancy
* Should have screening plasma HIV 1 RNA levels of 1000 c/mL to <=100,000 c/mL. If an independent review of accumulated data from other clinical trials investigating the DTG plus 3TC dual regimen is supportive of the DTG plus 3TC treatment regimen, enrolment will be opened to participants with Screening plasma HIV 1 RNA of 1000 c/mL to <=500,000 c/mL
* Participant should be antiretroviral naïve (defined as <=10 days of prior therapy with any antiretroviral agent following a diagnosis of HIV 1 infection). Participants who received HIV post exposure prophylaxis (PEP) or pre exposure prophylaxis (PrEP) in the past are allowed as long as the last PEP/PrEP dose was >1 year from HIV diagnosis or there is documented HIV seronegativity between the last prophylactic dose and the date of HIV diagnosis
* Participants or the participants legal representative capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and the protocol
* Participants enrolled in France: a participant will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category

Exclusion Criteria

* Women who are breastfeeding or plan to become pregnant or breastfeed during the study
* Any evidence of an active centers for disease control and prevention (CDC) Stage 3 disease (CDC, 2014), except cutaneous Kaposi's sarcoma not requiring systemic therapy and historical or current CD4 cell counts less than 200 cells/mm^3
* Participants with severe hepatic impairment (Class C) as determined by Child Pugh classification
* Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, oesophageal or gastric varices, or persistent jaundice), cirrhosis, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones
* Evidence of hepatitis B virus (HBV) infection or HBV surface antibody (anti-HBs or HBsAb) based on:

Participants positive for HBV surface antigen (HBsAg) at screening will be excluded Participants negative for HBV core antibody (anti HBs) but positive for anti HBc (negative HBsAg status) and positive for HBV deoxyribose nucleic acid (DNA) will be excluded; however, participants positive for anti HBc (negative HBsAg status) and positive for anti HBs (past and/or current evidence) are immune to HBV and will not be excluded

* Anticipated need for any hepatitis C virus (HCV) therapy during the first 48 weeks of the study and for HCV therapy based on interferon or any drugs that have a potential for adverse drug:drug interactions with study treatment throughout the entire study period
* Untreated syphilis infection positive RPR at Screening without clear documentation of treatment. Participants who are at least 14 days post completed treatment are eligible
* History or presence of allergy or intolerance to the study drugs or their components or drugs of their class
* Ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non invasive cutaneous squamous cell carcinoma, or cervical, anal or penile intraepithelial neoplasia; other localised malignancies require agreement between the investigator and the Study Medical Monitor for inclusion of the participant
* Participants who in the Investigator's judgment, poses a significant suicidality risk. Recent history of suicidal behaviour and/or suicidal ideation may be considered as evidence of serious suicide risk
* Treatment with an HIV 1 immunotherapeutic vaccine within 90 days of Screening
* Treatment with any of the following agents within 28 days of Screening:

  * Radiation therapy,
  * Cytotoxic chemotherapeutic agents,
  * Any systemic immune suppressant
* Treatment with any agent, except recognised ART as allowed above, with documented activity against HIV 1 in vitro within 28 days of first dose of study treatment
* Exposure to an experimental drug or experimental vaccine within either 28 days, 5 half lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is longer, prior to the first dose of study treatment
* Participants enrolled in France: the participant has participated in any study using an investigational drug during the previous 60 days or 5 half lives, or twice the duration of the biological effect of the experimental drug or vaccine, whichever is longer, prior to screening for the study or the participant will participate simultaneously in another clinical study
* Any evidence of pre existing viral resistance based on the presence of any major resistance associated mutation in the Screening result or, if known, in any historical resistance test result
* Any verified Grade 4 laboratory abnormality. A single repeat test is allowed during the Screening period to verify a result
* Any acute laboratory abnormality at Screening, which, in the opinion of the Investigator, would preclude the participants participation in the study of an investigational compound
* Alanine aminotransferase (ALT) >=5 times the upper limit of normal (ULN) or ALT >=3xULN and bilirubin >=1.5xULN (with >35% direct bilirubin)
* Creatinine clearance of <50 mL/min per 1.73 m^2 via the chronic kidney disease epidemiology collaboration (CKD EPI) method

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 722 (Actual)
Dates: Start 2016-07-18 (Actual); Primary Completion 2018-04-04 (Actual); Study Completion 2022-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (89):
- United States (23):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, San Leandro, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Ft. Pierce, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Berkley, Michigan
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Hillsborough, New Jersey
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
- Argentina (3):
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Córdoba
- Australia (5):
  - GSK Investigational Site, Darlinghurst, New South Wales
  - GSK Investigational Site, Parramatta, New South Wales
  - GSK Investigational Site, Fitzroy North, Victoria
  - GSK Investigational Site, Melbourne, Victoria
  - GSK Investigational Site, Prahran, Victoria
- Belgium (3):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Lodelinsart
- Canada (3):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- France (3):
  - GSK Investigational Site, Bobigny
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Paris
- Germany (5):
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Frankfurt am Main
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, München
- Italy (7):
  - GSK Investigational Site, Modena, Emilia-Romagna
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Turin, Piedmont
  - GSK Investigational Site, Bergamo
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Monza
- Mexico (3):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Distrito Federal
  - GSK Investigational Site, México
- GSK Investigational Site, Lima, Peru
- GSK Investigational Site, Bydgoszcz, Poland
- Portugal (3):
  - GSK Investigational Site, Amadora
  - GSK Investigational Site, Lisbon
  - GSK Investigational Site, Porto
- Romania (2):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Iași
- Russia (6):
  - GSK Investigational Site, Izhevsk
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Krasnodar
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, St.Peterburg
- Spain (8):
  - GSK Investigational Site, Alcorcón
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Marid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
- Switzerland (3):
  - GSK Investigational Site, Bern
  - GSK Investigational Site, Geneva
  - GSK Investigational Site, Zurich
- Taiwan (5):
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, New Taipei City
  - GSK Investigational Site, Tainan
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan District
- United Kingdom (5):
  - GSK Investigational Site, Woolwich, London, London
  - GSK Investigational Site, Brighton
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on ViiV's data sharing criteria can be found at: https://viivhealthcare.com/about-viiv/corporate-ethics-compliance/commitment-to-data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD is made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://viivhealthcare.com/about-viiv/corporate-ethics-compliance/commitment-to-data-transparency/

REFERENCES:
- [Background] Cahn P, Madero JS, Arribas JR, Antinori A, Ortiz R, Clarke AE, Hung CC, Rockstroh JK, Girard PM, Sievers J, Man C, Currie A, Underwood M, Tenorio AR, Pappa K, Wynne B, Fettiplace A, Gartland M, Aboud M, Smith K; GEMINI Study Team. Dolutegravir plus lamivudine versus dolutegravir plus tenofovir disoproxil fumarate and emtricitabine in antiretroviral-naive adults with HIV-1 infection (GEMINI-1 and GEMINI-2): week 48 results from two multicentre, double-blind, randomised, non-inferiority, phase 3 trials. Lancet. 2019 Jan 12;393(10167):143-155. doi: 10.1016/S0140-6736(18)32462-0. Epub 2018 Nov 9. PMID 30420123
- [Derived] Rolle CP, Arribas JR, Ortiz R, Underwood M, Parry CM, Grove R, DiMondi VP, Jones B, Kisare M. Efficacy and Safety Outcomes in Adults Initiating Dolutegravir/Lamivudine With High Viral Load in the GEMINI-1/-2 and STAT Trials. Open Forum Infect Dis. 2025 Mar 7;12(3):ofaf135. doi: 10.1093/ofid/ofaf135. eCollection 2025 Mar. PMID 40134635
- [Derived] Ait-Khaled M, Sierra Madero J, Estrada V, Gulminetti R, Hagins D, Tsai HC, Man C, Sievers J, Grove R, Zolopa A, Wynne B, van Wyk J. Impact of treatment adherence on efficacy of dolutegravir plus lamivudine and dolutegravir plus tenofovir disoproxil fumarate/emtricitabine: pooled analysis of the GEMINI-1 and GEMINI-2 clinical studies. HIV Res Clin Pract. 2021 Dec 9;23(1):9-14. Epub 2021 Dec 16. PMID 34913844

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study is a Phase 3, randomized, double-blind, parallel group, non-inferiority study. The study consisted of double-blind phase, open-label phase and continuation phase.
Pre-assignment Details: Total of 722 participants were enrolled and randomized; however only 719 participants (3 participants were never dosed following randomization) were dosed in to the study to receive either dolutegravir plus lamivudine (DTG+3TC) or dolutegravir plus tenofovir/emtricitabine (DTG+TDF/FTC) creating the intent to treat-exposed (ITT-E) Population.
Groups:
- DTG + 3TC - Double-blind Phase: Participants received a two-drug regimen of DTG + 3TC administered orally, once daily for 96 weeks in a double-blind phase.
- DTG + TDF/FTC - Double-blind Phase: Participants received a three-drug regimen of DTG + TDF/FTC fixed dose combination (FDC) administered orally, once daily for 96 weeks in a double-blind phase.
- DTG + 3TC - Open-label Phase: Participants received a two-drug regimen of DTG + 3TC administered orally, once daily from Week 96 to Week 148 in an open-label phase.
- DTG + TDF/FTC - Open-label Phase: Participants received a three-drug regimen of DTG + TDF/FTC FDC administered orally, once daily from Week 96 to Week 148 in an open-label phase.
- DTG + 3TC - Continuation Phase: Participants received a DTG + 3TC administered orally, once daily from Week 148 to Week 280 in a continuation phase.
Period: Double-blind Phase (Day1 to Week 96)
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase | DTG + 3TC - Open-label Phase | DTG + TDF/FTC - Open-label Phase | DTG + 3TC - Continuation Phase
Started | 360 (Randomized) | 362 (Randomized) | 0 | 0 | 0
Intent-to-Treat Exposed | 360 | 359 | 0 | 0 | 0
Completed | 319 | 327 | 0 | 0 | 0
Not Completed | 41 | 35 | 0 | 0 | 0
Not completed — Protocol specific withdrawal criteria | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 9 | 0 | 0 | 0
Not completed — Physician Decision | 3 | 3 | 0 | 0 | 0
Not completed — Lost to Follow-up | 9 | 7 | 0 | 0 | 0
Not completed — Adverse Event | 10 | 6 | 0 | 0 | 0
Not completed — Lack of Efficacy | 5 | 2 | 0 | 0 | 0
Not completed — Protocol Deviation | 5 | 3 | 0 | 0 | 0
Not completed — Randomized, but did not receive treatment | 0 | 3 | 0 | 0 | 0
Period: Open-label Phase (Week 96 to Week 148)
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase | DTG + 3TC - Open-label Phase | DTG + TDF/FTC - Open-label Phase | DTG + 3TC - Continuation Phase
Started | 0 | 0 | 319 | 327 | 0
Completed | 0 | 0 | 301 | 300 | 0
Not Completed | 0 | 0 | 18 | 27 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 6 | 0
Not completed — Lack of Efficacy | 0 | 0 | 2 | 0 | 0
Not completed — Protocol Deviation | 0 | 0 | 2 | 2 | 0
Not completed — Protocol-Specified Withdrawal Criteria | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 4 | 7 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 7 | 9 | 0
Period: Continuation Phase(Week 148 to Week 280)
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase | DTG + 3TC - Open-label Phase | DTG + TDF/FTC - Open-label Phase | DTG + 3TC - Continuation Phase
Started | 0 | 0 | 0 | 0 | 252 (252 participants from the Open-label Phase entered in the Continuation Phase)
Completed | 0 | 0 | 0 | 0 | 239
Not Completed | 0 | 0 | 0 | 0 | 13
Not completed — Protocol Deviation | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 5

BASELINE CHARACTERISTICS:
Population: Baseline Characteristic data are reported for the Intent-to-Treat Exposed (ITT-E) Population consisted of all randomized participants who received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase | Total
Number analyzed (Participants) | 360 | 359 | 719
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.6 (10.72) | 34.4 (10.35) | 34.5 (10.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 46 | 100
  Male | 306 | 313 | 619
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American (Am) Indian or Alaska (Al.) native | 21 | 29 | 50
  Asian-Central/South Asian heritage (H.) | 0 | 3 | 3
  Asian - East Asian H. | 28 | 26 | 54
  Asian - South East Asian H. | 6 | 1 | 7
  Black or African Am | 51 | 35 | 86
  Native Hawaiian or other Pacific Islander | 0 | 1 | 1
  White (Wt)-Arabic/North African H. | 3 | 3 | 6
  Wt-Wt/Caucasian (Ca.)/European (Eu.) H. | 237 | 249 | 486
  Multiple | 14 | 12 | 26

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Plasma Human Immunodeficiency Virus Type 1 (HIV-1) Ribonucleic Acid (RNA) <50 Copies/mL (c/mL) at Week 48
Description: Percentage of participants with HIV-1 RNA<50 c/mL was obtained using Food and Drug Administration (FDA) Snapshot algorithm. The Snapshot algorithm treated all participants without HIV-1 RNA data at the visit of interest (due to missing data or discontinuation of investigational product prior to the visit window) as non-responders, as well as participants who switch their concomitant antiretroviral therapy (ART) prior to the visit of interest. This endpoint was analyzed using a stratified analysis with Cochran-Mantel-Haenszel (CMH) weights. Intent-To-Treat Exposed (ITT-E) Population was used which comprised of all randomized participants who received at least one dose of study treatment. Percentage values are rounded off.
Time Frame: Week 48
Population: ITT-E Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 360 | 359
Percentage of participants | 93 [90.4 to 95.7] | 94 [91.4 to 96.4]
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Non-Inferiority — Treatment with DTG+ 3TC was to be declared non-inferior to treatment with DTG+TDF/FTC if the lower end of a two-sided 95% confidence interval for the difference between the two groups in response rates at Week 48 was greater than -10%; Adjusted difference in proportion = -0.7, 95% CI 2-sided [-4.3 to 2.9] — Difference in proportion was based on CMH stratified analysis adjusting for Baseline stratification factors: Plasma HIV-1 RNA (<= vs. >100,000 copies per milliliter) and CD4+ cell count (<= vs. >200 cells per cubic millimeter [cells/mm^3])

2. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 c/mL at Week 24
Description: Percentage of participants with HIV-1 RNA<50 c/mL was obtained using FDA Snapshot algorithm. The Snapshot algorithm treated all participants without HIV-1 RNA data at the visit of interest (due to missing data or discontinuation of investigational product prior to the visit window) as non-responders, as well as participants who switch their concomitant ART prior to the visit of interest. This endpoint was analyzed using a stratified analysis with CMH weights. Percentage values are rounded off.
Time Frame: Week 24
Population: ITT-E Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 360 | 359
Percentage of participants | 94 [91.4 to 96.4] | 94 [91.4 to 96.4]
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Non-Inferiority — Treatment with DTG+ 3TC was to be declared non-inferior to treatment with DTG+TDF/FTC if the lower end of a two-sided 95% confidence interval for the difference between the two groups in response rates at Week 24 was greater than -10%; Adjusted difference in proportion = 0.1, 95% CI 2-sided [-3.4 to 3.6] — Difference in proportion was based on CMH stratified analysis adjusting for Baseline stratification factors: Plasma HIV-1 RNA (<= vs. >100,000 c/mL) and CD4+ cell count (<= vs. >200 cells/mm^3)

3. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 c/mL at Week 96
Description: as for outcome 2
Time Frame: Week 96
Population: ITT-E Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 360 | 359
Percentage of participants | 88 [84.4 to 91.2] | 90 [86.5 to 92.8]
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Adjusted difference in proportion = -1.8, 95% CI 2-sided [-6.4 to 2.7] — Week 96. Difference in proportion was based on CMH stratified analysis adjusting for Baseline stratification factors: Plasma HIV-1 RNA (<= vs. >100,000 c/mL) and CD4+ cell count (<= vs. >200 cells/mm^3)

4. Secondary Outcome: Percentage of Participants With Plasma HIV-1 RNA <50 c/mL at Week 144
Description: as for outcome 2
Time Frame: Week 144
Population: ITT-E Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- DTG + 3TC - Double-blind Phase + Open-label Phase: Participants received a two-drug regimen of DTG + 3TC administered orally, once daily until Week 96 in double-blind phase and participants continued to receive DTG + 3TC from Week 96 to Week 148 in an open-label phase.
- DTG + TDF/FTC - Double-blind Phase + Open-label Phase: Participants received a three-drug regimen of DTG + TDF/FTC FDC administered orally, once daily until Week 96 in double-blind phase and participants continued to receive DTG + TDF/FTC FDC from Week 96 to Week 148 in an open-label phase.
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 360 | 359
Percentage of participants | 84 [80.4 to 87.9] | 84 [80.6 to 88.2]
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; Adjusted difference in proportion = 0.0, 95% CI 2-sided [-5.3 to 5.3] — Week 144. Difference in proportion was based on CMH stratified analysis adjusting for Baseline stratification factors: Plasma HIV-1 RNA (<= vs. >100,000 c/mL) and CD4+ cell count (<= vs. >200 cells/mm^3)

5. Secondary Outcome: Time to Viral Suppression (HIV-1 RNA <50 c/mL) up to Week 144
Description: Time of viral suppression is defined as the first viral load value <50 c/mL. Nonparametric Kaplan-Meier method was performed. Participants who withdrew for any reason without being suppressed were censored at date of withdrawal. Participants who have not been withdrawn and have not had viral suppression at time of the analysis were censored at last viral load date. Confidence Interval (CI) was estimated using the Brookmeyer-Crowley method.
Time Frame: Up to Week 144
Population: ITT-E Population
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 360 | 359
Days | 29.0 [29.0 to 55.0] | 29.0 [29.0 to 57.0]
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; p = 0.797, Generalised Wilcoxon procedure — The generalised Wilcoxon procedure was used to estimate a p-value for detecting a difference in cumulative incidence curves between treatment groups; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.88 to 1.19] — Hazard ratios were estimated using the Cox proportional hazard regression model

6. Secondary Outcome: CD4+ Cell Counts at Weeks 24 and 48
Description: CD4+ cells are type of white blood cells that fight infection and as HIV infection progresses, the number of these cells declines. Blood samples were collected at specified time points to assess CD4+ cells. Analysis was performed by flow cytometry.
Time Frame: Weeks 24 and 48
Population: ITT-E Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Cells/mm^3
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 360 | 359
Cells/mm^3
  Week 24, n=349,345: number analyzed (Participants) | 349 | 345
  Week 24, n=349,345 | 650.4 (257.02) | 633.0 (287.37)
  Week 48, n=337,340: number analyzed (Participants) | 337 | 340
  Week 48, n=337,340 | 688.1 (266.39) | 689.8 (308.49)

7. Secondary Outcome: CD4+ Cell Counts at Week 96
Description: as for outcome 6
Time Frame: Week 96
Population: ITT-E Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Cells/mm^3
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 318 | 327
Cells/mm^3 | 734.9 (270.82) | 739.9 (299.80)

8. Secondary Outcome: CD4+ Cell Counts at Week 144
Description: as for outcome 6
Time Frame: Week 144
Population: ITT-E Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Cells/mm^3
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 296 | 292
Cells/mm^3 | 763.8 (266.61) | 770.4 (332.65)

9. Secondary Outcome: Changes From Baseline in CD4+ Cell Counts at Week 24 and 48
Description: CD4+ cells are type of white blood cells that fight infection and as HIV infection progresses, the number of these cells declines. Blood samples were collected at specified time points to assess CD4+ cells. Analysis was performed by flow cytometry. Baseline value is defined as the the latest pre-dose assessment. Change from Baseline was defined as value at the indicated time point minus Baseline value. Adjusted least mean and standard error has been presented. Adjusted mean is the estimated mean change from Baseline at each visit in each arm calculated from a repeated measures model adjusting for the following covariates/factors: treatment, visit, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, treatment and visit interaction, and Baseline CD4+ cell count and visit interaction, with visit as the repeated factor.
Time Frame: Baseline and Weeks 24, 48
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Cells/mm^3
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 360 | 359
Cells/mm^3
  Week 24, n=349, 345: number analyzed (Participants) | 349 | 345
  Week 24, n=349, 345 | 188.8 (8.77) | 163.2 (9.08)
  Week 48, n=337, 340: number analyzed (Participants) | 337 | 340
  Week 48, n=337, 340 | 225.7 (8.94) | 217.2 (9.93)
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p = 0.043, Mixed Model Repeated Measures (MMRM); Mean Difference (Net) = 25.6, 95% CI 2-sided [0.8 to 50.4] — Week 24. Following covariates/factors were adjusted: treatment, visit, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, treatment and visit interaction and Baseline CD4+ cell count and visit interaction with visit as the repeated factor
Statistical Analysis 2: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p = 0.523, MMRM; Mean Difference (Net) = 8.5, 95% CI 2-sided [-17.7 to 34.8] — Week 48. Following covariates/factors were adjusted: treatment, visit, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, treatment and visit interaction and Baseline CD4+ cell count and visit interaction with visit as the repeated factor

10. Secondary Outcome: Changes From Baseline in CD4+ Cell Counts at Week 96
Description: CD4+ cells are type of white blood cells that fight infection and as HIV infection progresses, the number of these cells declines. Blood samples were collected at specified time points to assess CD4+ cells. Analysis was performed by flow cytometry. Baseline value is defined as the the latest pre-dose assessment. Change from Baseline was defined as value at the indicated time point minus Baseline value. Adjusted mean and standard error has been presented. Adjusted mean is the estimated mean change from Baseline at each visit in each arm calculated from a repeated measures model adjusting for the following covariates/factors: treatment, visit, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, treatment and visit interaction, and Baseline CD4+ cell count and visit interaction, with visit as the repeated factor.
Time Frame: Baseline and Week 96
Population: ITT-E Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Cells/mm^3
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 318 | 327
Cells/mm^3 | 272.0 (10.83) | 264.6 (11.18)
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p = 0.635, Mixed Model Repeated Measures (MMRM); Mean Difference (Net) = 7.4, 95% CI 2-sided [-23.2 to 38.0] — Week 96. Following covariates/factors were adjusted: treatment, visit, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, treatment and visit interaction and Baseline CD4+ cell count and visit interaction with visit as the repeated factor

11. Secondary Outcome: Changes From Baseline in CD4+ Cell Counts at Week 144
Description: as for outcome 10
Time Frame: Baseline and Week 144
Population: ITT-E Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Cells/mm^3
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 296 | 292
Cells/mm^3 | 301.7 (11.55) | 296.6 (13.55)
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; p = 0.777, MMRM; Mean Difference (Net) = 5.1, 95% CI 2-sided [-29.9 to 40.0] — Week 144.Following covariates/factors were adjusted: treatment, visit, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, treatment and visit interaction and Baseline CD4+ cell count and visit interaction with visit as the repeated factor

12. Secondary Outcome: Number of Participants With HIV-1 Disease Progression up to Week 144
Description: HIV-associated conditions were recorded during the study and was assessed according to the 2014 Centers for Disease Control and Prevention (CDC) Classification System for HIV Infection in Adults. Disease progressions summarize participants who had HIV infection stage 3 associated conditions or death. Indicators of clinical disease progression were defined as: CDC Category Stage 1 at enrollment to Stage 3 event; CDC Category Stage 2 at enrolment to Stage 3 event; CDC Category Stage 3 at enrollment to New Stage 3 Event; CDC Category Stage 1, 2 or 3 at enrolment to Death. Participants may have more than one indicators of clinical disease progression including death, hence they may contribute to data in more than one categories.
Time Frame: Up to Week 144
Population: ITT-E Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 360 | 359
Participants
  No disease progression | 356 | 357
  From CDC Stage 1 to CDC Stage 3 Event | 0 | 0
  From CDC Stage 2 to CDC Stage 3 Event | 2 | 1
  From CDC Stage 3 to New CDC Stage 3 Event | 1 | 0
  From CDC Stage 1, 2 or 3 to Death | 2 | 1

13. Secondary Outcome: Number of Participants With Treatment-emergent Genotypic Resistance up to Week 144
Description: Number of participants, who met confirmed virologic withdrawal (CVW) criteria, with treatment emergent genotypic resistance to Integrase strand transfer inhibitor (INSTI) and/or Nucleoside reverse transcriptase inhibitor (NRTI) was summarized. The Viral Genotypic Population comprised of all participants in the ITT-E population who have available on-treatment genotypic resistance data.
Time Frame: Up to Week 144
Population: Viral Genotypic Population. Only those participants available at the specified time points were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 7 | 3
Participants
  INSTI Mutations | 0 | 0
  Major mutations of the NRTI | 0 | 0

14. Secondary Outcome: Number of Participants With Treatment-emergent Phenotypic Resistance up to Week 144
Description: Number of participants, who met CVW criteria, with treatment emergent phenotypic resistance to INSTI and/or NRTI were summarized. Assessment of antiviral activity of anti-retroviral therapy (ART) using phenotypic test results were interpreted through a proprietary algorithm (from Monogram Biosciences) and provides the overall susceptibility of the drugs (DTG, 3TC, Abacavir [ABC], elvitegravir [EGV], raltegravir [RAL], zidovudine [AZT], stavudine [D4T], didanosine [DDI]), emtricitabine [FTC], tenofovir disiproxil fumarate [TDF]). Partially sensitive and resistant cells were considered resistant in this analysis. The Viral Phenotypic Population comprised of all participants in the ITT-E population who have available on-treatment phenotypic resistance data.
Time Frame: Up to Week 144
Population: Viral Phenotypic Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 7 | 4
Participants
  INSTI, DTG, Sensitive, n=7,2: number analyzed (Participants) | 7 | 2
  INSTI, DTG, Sensitive, n=7,2 | 7 | 2
  INSTI, DTG, Resistant, n=7,2: number analyzed (Participants) | 7 | 2
  INSTI, DTG, Resistant, n=7,2 | 0 | 0
  INSTI, EGV, Sensitive, n=7,2: number analyzed (Participants) | 7 | 2
  INSTI, EGV, Sensitive, n=7,2 | 7 | 2
  INSTI, EGV, Resistant, n=7,2: number analyzed (Participants) | 7 | 2
  INSTI, EGV, Resistant, n=7,2 | 0 | 0
  INSTI, RAL, Sensitive, n=7,2: number analyzed (Participants) | 7 | 2
  INSTI, RAL, Sensitive, n=7,2 | 7 | 2
  INSTI, RAL, Resistant, n=7,2: number analyzed (Participants) | 7 | 2
  INSTI, RAL, Resistant, n=7,2 | 0 | 0
  NRTI, 3TC, Sensitive, n=7,3: number analyzed (Participants) | 7 | 3
  NRTI, 3TC, Sensitive, n=7,3 | 7 | 3
  NRTI, 3TC, Resistant, n=7,3: number analyzed (Participants) | 7 | 3
  NRTI, 3TC, Resistant, n=7,3 | 0 | 0
  NRTI, ABC, Sensitive, n=7,3: number analyzed (Participants) | 7 | 3
  NRTI, ABC, Sensitive, n=7,3 | 7 | 3
  NRTI, ABC, Resistant, n=7,3: number analyzed (Participants) | 7 | 3
  NRTI, ABC, Resistant, n=7,3 | 0 | 0
  NRTI, AZT, Sensitive, n=7,3: number analyzed (Participants) | 7 | 3
  NRTI, AZT, Sensitive, n=7,3 | 7 | 3
  NRTI, AZT, Resistant, n=7,3: number analyzed (Participants) | 7 | 3
  NRTI, AZT, Resistant, n=7,3 | 0 | 0
  NRTI, D4T, Sensitive, n=7,3: number analyzed (Participants) | 7 | 3
  NRTI, D4T, Sensitive, n=7,3 | 7 | 3
  NRTI, D4T, Resistant, n=7,3: number analyzed (Participants) | 7 | 3
  NRTI, D4T, Resistant, n=7,3 | 0 | 0
  NRTI, DDI, Sensitive, n=7,3: number analyzed (Participants) | 7 | 3
  NRTI, DDI, Sensitive, n=7,3 | 7 | 3
  NRTI, DDI, Resistant, n=7,3: number analyzed (Participants) | 7 | 3
  NRTI, DDI, Resistant, n=7,3 | 0 | 0
  NRTI, FTC, Sensitive, n=7,3: number analyzed (Participants) | 7 | 3
  NRTI, FTC, Sensitive, n=7,3 | 7 | 3
  NRTI, FTC, Resistant, n=7,3: number analyzed (Participants) | 7 | 3
  NRTI, FTC, Resistant, n=7,3 | 0 | 0
  NRTI, TDF, Sensitive, n=7,3: number analyzed (Participants) | 7 | 3
  NRTI, TDF, Sensitive, n=7,3 | 7 | 3
  NRTI, TDF, Resistant, n=7,3: number analyzed (Participants) | 7 | 3
  NRTI, TDF, Resistant, n=7,3 | 0 | 0

15. Secondary Outcome: Number of Participants With Any Adverse Event (AE) and Serious AE (SAE) up to Week 148
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention or protocol-defined event associated with liver injury and impaired liver function were categorized as SAE. Safety Population was used which comprised of all participants who received at least one dose of study treatment.
Time Frame: Up to Week 148
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 360 | 359
Participants
  Any AE | 306 | 309
  Any SAE | 39 | 47

16. Secondary Outcome: Number of Participants With AEs by Maximum Severity Grades up to Week 148
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AEs were evaluated by the investigator and graded according to the Division of Acquired Immunodeficiency Syndrome (DAIDS) toxicity scales from Grade 1 to 5 (1=Mild, 2=Moderate, 3=Severe, 4=Potentially life threatening, 5=Death). The higher the grade, the more severe the symptoms. Number of participants with adverse events by maximum grade have been presented.
Time Frame: Up to Week 148
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 360 | 359
Participants
  Grade 1 AEs | 54 | 54
  Grade 2 AEs | 211 | 205
  Grade 3 AEs | 32 | 43
  Grade 4 AEs | 7 | 6
  Grade 5 AEs | 2 | 1

17. Secondary Outcome: Number of Participants With Any Drug Related AEs and Drug Related AEs by Maximum Grade up to Week 148
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AEs were evaluated by the investigator and graded according to the DAIDS toxicity scales from Grade 1 to 5. (1=Mild, 2=Moderate, 3=Severe, 4=Potentially life threatening, 5=Death). The higher the grade, the more severe the symptoms. Number of participants with drug related AEs and drug related AEs by by maximum grade have been presented.
Time Frame: Up to Week 148
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 360 | 359
Participants
  Any drug related AE | 69 | 91
  Drug related AEs with maximum toxicity Grade 1 | 37 | 53
  Drug related AEs with maximum toxicity Grade 2 | 26 | 29
  Drug related AEs with maximum toxicity Grade 3 | 5 | 8
  Drug related AEs with maximum toxicity Grade 4 | 1 | 1
  Drug related AEs with maximum toxicity Grade 5 | 0 | 0

18. Secondary Outcome: Number of Participants With Maximum Post-Baseline Emergent Hematology Toxicities up to Week 144
Description: Blood samples were collected up to Week 144 for assessment of hemoglobin, leukocytes, neutrophils and platelet count. Any abnormality was graded according to DAIDS toxicity scales from Grade 1 to 4 (1=Mild, 2=Moderate, 3=Severe, 4=Potentially life threatening). The higher the grade, the more severe the symptoms. Only those participants with maximum post-Baseline emergent hematology toxicities in any of the listed hematology parameters have been presented.
Time Frame: Up to Week 144
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 360 | 359
Participants
  Hemoglobin, Grades 1 to 4 | 8 | 10
  Hemoglobin, Grades 2 to 4 | 6 | 6
  Hemoglobin, Grades 3 to 4 | 2 | 1
  Hemoglobin, Grade 1 | 2 | 4
  Hemoglobin, Grade 2 | 4 | 5
  Hemoglobin, Grade 3 | 1 | 1
  Hemoglobin, Grade 4 | 1 | 0
  Leukocytes, Grades 1 to 4 | 5 | 5
  Leukocytes, Grades 2 to 4 | 1 | 0
  Leukocytes, Grades 3 to 4 | 0 | 0
  Leukocytes, Grade 1 | 4 | 5
  Leukocytes, Grade 2 | 1 | 0
  Leukocytes, Grade 3 | 0 | 0
  Leukocytes, Grade 4 | 0 | 0
  Neutrophils, Grades 1 to 4 | 23 | 7
  Neutrophils, Grades 2 to 4 | 8 | 3
  Neutrophils, Grades 3 to 4 | 4 | 1
  Neutrophils, Grade 1 | 15 | 4
  Neutrophils, Grade 2 | 4 | 2
  Neutrophils, Grade 3 | 2 | 1
  Neutrophils, Grade 4 | 2 | 0
  Platelets, Grades 1 to 4 | 13 | 9
  Platelets, Grades 2 to 4 | 5 | 5
  Platelets, Grades 3 to 4 | 0 | 0
  Platelets, Grade 1 | 8 | 4
  Platelets, Grade 2 | 5 | 5
  Platelets, Grade 3 | 0 | 0
  Platelets, Grade 4 | 0 | 0

19. Secondary Outcome: Number of Participants With Maximum Post-Baseline Emergent Chemistry Toxicities up to Week 144
Description: Blood samples were collected up to Week 144 for assessment of Alanine Aminotransferase (ALT), Albumin, Alkaline Phosphatase (ALP), Aspartate aminotransferase (AST), Bilirubin, Carbon dioxide (CO2), Cholesterol, Creatine kinase (CK), Creatinine, Direct Bilirubin, Glomerular filtration rate (GFR), Hypercalcemia, Hyperglycemia, Hyperkalemia, Hypernatremia, Hypocalcemia, Hypoglycemia, Hypokalemia, Hyponatremia, Low density lipid (LDL) Cholesterol, Lactate Dehydrogenase, Lipase, Phosphate, and Triglycerides. Any abnormality was graded according to DAIDS toxicity scales from Grade 1 to 4 (1=Mild, 2=Moderate, 3=Severe, 4=Potentially life threatening). The higher the grade, the more severe the symptoms. Only those participants with maximum post-Baseline emergent chemistry toxicities in any of the chemistry parameters have been presented.
Time Frame: Up to Week 144
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 360 | 359
Participants
  ALT, Grades 1 to 4 | 77 | 71
  ALT, Grades 2 to 4 | 30 | 29
  ALT, Grades 3 to 4 | 13 | 15
  ALT, Grade 1 | 47 | 42
  ALT, Grade 2 | 17 | 14
  ALT, Grade 3 | 6 | 8
  ALT, Grade 4 | 7 | 7
  Albumin, Grades 1 to 4 | 2 | 1
  Albumin, Grades 2 to 4 | 2 | 1
  Albumin, Grades 3 to 4 | 0 | 1
  Albumin, Grade 1 | 0 | 0
  Albumin, Grade 2 | 2 | 0
  Albumin, Grade 3 | 0 | 1
  Albumin, Grade 4 | 0 | 0
  ALP, Grades 1 to 4 | 10 | 17
  ALP, Grades 2 to 4 | 2 | 3
  ALP, Grades 3 to 4 | 0 | 1
  ALP, Grade 1 | 8 | 14
  ALP, Grade 2 | 2 | 2
  ALP, Grade 3 | 0 | 1
  ALP, Grade 4 | 0 | 0
  AST, Grades 1 to 4 | 71 | 83
  AST, Grades 2 to 4 | 30 | 32
  AST, Grades 3 to 4 | 15 | 14
  AST, Grade 1 | 41 | 51
  AST, Grade 2 | 15 | 18
  AST, Grade 3 | 8 | 11
  AST, Grade 4 | 7 | 3
  Bilirubin, Grades 1 to 4 | 46 | 56
  Bilirubin, Grades 2 to 4 | 13 | 16
  Bilirubin, Grades 3 to 4 | 4 | 3
  Bilirubin, Grade 1 | 33 | 40
  Bilirubin, Grade 2 | 9 | 13
  Bilirubin, Grade 3 | 0 | 2
  Bilirubin, Grade 4 | 4 | 1
  CO2, Grades 1 to 4 | 111 | 111
  CO2, Grades 2 to 4 | 10 | 4
  CO2, Grades 3 to 4 | 0 | 0
  CO2, Grade 1 | 101 | 107
  CO2, Grade 2 | 10 | 4
  CO2, Grade 3 | 0 | 0
  CO2, Grade 4 | 0 | 0
  Cholesterol, Grades 1 to 4 | 98 | 50
  Cholesterol, Grades 2 to 4 | 23 | 12
  Cholesterol, Grades 3 to 4 | 1 | 0
  Cholesterol, Grade 1 | 75 | 38
  Cholesterol, Grade 2 | 22 | 12
  Cholesterol, Grade 3 | 1 | 0
  Cholesterol, Grade 4 | 0 | 0
  CK, Grades 1 to 4 | 91 | 83
  CK, Grades 2 to 4 | 49 | 47
  CK, Grades 3 to 4 | 29 | 28
  CK, Grade 1 | 42 | 36
  CK, Grade 2 | 20 | 19
  CK, Grade 3 | 11 | 11
  CK, Grade 4 | 18 | 17
  Creatinine, Grades 1 to 4 | 18 | 28
  Creatinine, Grades 2 to 4 | 5 | 2
  Creatinine, Grades 3 to 4 | 0 | 1
  Creatinine, Grade 1 | 13 | 26
  Creatinine, Grade 2 | 5 | 1
  Creatinine, Grade 3 | 0 | 1
  Creatinine, Grade 4 | 0 | 0
  Direct Bilirubin, Grades 1 to 4 | 11 | 10
  Direct Bilirubin, Grades 2 to 4 | 11 | 10
  Direct Bilirubin, Grades 3 to 4 | 11 | 10
  Direct Bilirubin, Grade 1 | 0 | 0
  Direct Bilirubin, Grade 2 | 0 | 0
  Direct Bilirubin, Grade 3 | 11 | 10
  Direct Bilirubin, Grade 4 | 0 | 0
  GFR, Grades 1 to 4 | 198 | 219
  GFR, Grades 2 to 4 | 198 | 219
  GFR, Grades 3 to 4 | 20 | 29
  GFR, Grade 1 | 0 | 0
  GFR, Grade 2 | 178 | 190
  GFR, Grade 3 | 20 | 28
  GFR, Grade 4 | 0 | 1
  Hypercalcaemia, Grades 1 to 4 | 4 | 5
  Hypercalcaemia, Grades 2 to 4 | 0 | 1
  Hypercalcaemia, Grades 3 to 4 | 0 | 1
  Hypercalcemia, Grade 1 | 4 | 4
  Hypercalcaemia, Grade 2 | 0 | 0
  Hypercalcaemia, Grade 3 | 0 | 0
  Hypercalcaemia, Grade 4 | 0 | 1
  Hyperglycaemia, Grades 1 to 4 | 106 | 86
  Hyperglycaemia, Grades 2 to 4 | 49 | 38
  Hyperglycaemia, Grades 3 to 4 | 3 | 3
  Hyperglycaemia, Grade 1 | 57 | 48
  Hyperglycaemia, Grade 2 | 46 | 35
  Hyperglycaemia, Grade 3 | 2 | 2
  Hyperglycaemia, Grade 4 | 1 | 1
  Hyperkalemia, Grades 1 to 4 | 7 | 7
  Hyperkalemia, Grades 2 to 4 | 2 | 1
  Hyperkalemia, Grades 3 to 4 | 1 | 1
  Hyperkalemia, Grade 1 | 5 | 6
  Hyperkalemia, Grade 2 | 1 | 0
  Hyperkalemia, Grade 3 | 0 | 1
  Hyperkalemia, Grade 4 | 1 | 0
  Hypernatremia, Grades 1 to 4 | 4 | 7
  Hypernatremia, Grades 2 to 4 | 1 | 0
  Hypernatremia, Grades 3 to 4 | 0 | 0
  Hypernatremia, Grade 1 | 3 | 7
  Hypernatremia, Grade 2 | 1 | 0
  Hypernatremia, Grade 3 | 0 | 0
  Hypernatremia, Grade 4 | 0 | 0
  Hypocalcaemia, Grades 1 to 4 | 17 | 21
  Hypocalcaemia, Grades 2 to 4 | 6 | 11
  Hypocalcaemia, Grades 3 to 4 | 1 | 3
  Hypocalcaemia, Grade 1 | 11 | 10
  Hypocalcaemia, Grade 2 | 5 | 8
  Hypocalcaemia, Grade 3 | 1 | 2
  Hypocalcaemia, Grade 4 | 0 | 1
  Hypoglycaemia, Grades 1 to 4 | 22 | 21
  Hypoglycaemia, Grades 2 to 4 | 6 | 5
  Hypoglycaemia, Grades 3 to 4 | 4 | 1
  Hypoglycaemia, Grade 1 | 16 | 16
  Hypoglycaemia, Grade 2 | 2 | 4
  Hypoglycaemia, Grade 3 | 3 | 0
  Hypoglycaemia, Grade 4 | 1 | 1
  Hypokalemia, Grades 1 to 4 | 9 | 5
  Hypokalemia, Grades 2 to 4 | 0 | 1
  Hypokalemia, Grades 3 to 4 | 0 | 0
  Hypokalemia, Grade 1 | 9 | 4
  Hypokalemia, Grade 2 | 0 | 1
  Hypokalemia, Grade 3 | 0 | 0
  Hypokalemia, Grade 4 | 0 | 0
  Hyponatremia, Grades 1 to 4 | 23 | 22
  Hyponatremia, Grades 2 to 4 | 0 | 3
  Hyponatremia, Grades 3 to 4 | 0 | 1
  Hyponatremia, Grade 1 | 23 | 19
  Hyponatremia, Grade 2 | 0 | 2
  Hyponatremia, Grade 3 | 0 | 0
  Hyponatremia, Grade 4 | 0 | 1
  LDL Cholesterol, Grades 1 to 4 | 66 | 40
  LDL Cholesterol, Grades 2 to 4 | 21 | 13
  LDL Cholesterol, Grades 3 to 4 | 6 | 2
  LDL Cholesterol, Grade 1 | 45 | 27
  LDL Cholesterol, Grade 2 | 15 | 11
  LDL Cholesterol, Grade 3 | 6 | 2
  LDL Cholesterol, Grade 4 | 0 | 0
  Lactate Dehydrogenase, Grades 1 to 4 | 4 | 2
  Lactate Dehydrogenase, Grades 2 to 4 | 3 | 0
  Lactate Dehydrogenase, Grades 3 to 4 | 0 | 0
  Lactate Dehydrogenase, Grade 1 | 1 | 2
  Lactate Dehydrogenase, Grade 2 | 3 | 0
  Lactate Dehydrogenase, Grade 3 | 0 | 0
  Lactate Dehydrogenase, Grade 4 | 0 | 0
  Lipase, Grades 1 to 4 | 72 | 81
  Lipase, Grades 2 to 4 | 37 | 43
  Lipase, Grades 3 to 4 | 9 | 17
  Lipase, Grade 1 | 35 | 38
  Lipase, Grade 2 | 28 | 26
  Lipase, Grade 3 | 6 | 13
  Lipase, Grade 4 | 3 | 4
  Phosphate, Grades 1 to 4 | 75 | 78
  Phosphate, Grades 2 to 4 | 50 | 51
  Phosphate, Grades 3 to 4 | 7 | 7
  Phosphate, Grade 1 | 25 | 27
  Phosphate, Grade 2 | 43 | 44
  Phosphate, Grade 3 | 7 | 7
  Phosphate, Grade 4 | 0 | 0
  Triglycerides, Grades 1 to 4 | 89 | 75
  Triglycerides, Grades 2 to 4 | 22 | 15
  Triglycerides, Grades 3 to 4 | 4 | 1
  Triglycerides, Grade 1 | 67 | 60
  Triglycerides, Grade 2 | 18 | 14
  Triglycerides, Grade 3 | 4 | 1
  Triglycerides, Grade 4 | 0 | 0

20. Secondary Outcome: Number of Participants Who Discontinue Treatment Due to AEs Over Weeks 24, 48, 96
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Number of participants who discontinued treatment due to AEs have been reported.
Time Frame: Up to Weeks 24, 48 and 96
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 360 | 359
Participants
  Week 24 | 6 | 4
  Week 48 | 8 | 8
  Week 96 | 10 | 12

21. Secondary Outcome: Number of Participants Who Discontinue Treatment Due to AEs Over Week 144
Description: as for outcome 20
Time Frame: Up to Week 144
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 360 | 359
Participants | 13 | 16

22. Secondary Outcome: Change From Baseline in Renal Biomarkers-Serum Cystatin C and Serum Retinol Binding Protein (RBP) at Weeks 24, 48
Description: Blood and/or urine samples were collected to perform evaluation of renal biomarkers which included Serum Cystatin C and Serum RBP. Baseline value is the latest pre-dose assessment. Change from Baseline was defined as value at indicated time point minus Baseline value. Biomarkers were adjusted for treatment, visit, Baseline plasma HIV-1 RNA, Baseline CD4+ cell count, age, sex, race, presence of diabetes mellitus, presence of hypertension, Baseline biomarker value, treatment and visit interaction, and Baseline biomarker value and visit interaction; with visit as the repeated factor.
Time Frame: Baseline and at Weeks 24, 48
Population: Safety Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Least Squares Mean (Standard Error); unit: Milligrams per Liter (mg/L)
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 360 | 359
Milligrams per Liter (mg/L)
  Serum Cystatin C, Week 24, n=345,345: number analyzed (Participants) | 345 | 345
  Serum Cystatin C, Week 24, n=345,345 | -0.04 (0.005) | 0.00 (0.005)
  Serum Cystatin C, Week 48, n=335,336: number analyzed (Participants) | 335 | 336
  Serum Cystatin C, Week 48, n=335,336 | -0.05 (0.005) | -0.04 (0.006)
  Serum RBP, Week 24, n=345,343: number analyzed (Participants) | 345 | 343
  Serum RBP, Week 24, n=345,343 | 1.2 (0.42) | 1.4 (0.48)
  Serum RBP, Week 48, n=334, 334: number analyzed (Participants) | 334 | 334
  Serum RBP, Week 48, n=334, 334 | 0.6 (0.45) | -0.1 (0.42)
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p < 0.001, MMRM; Mean Difference (Net) = -0.03, 95% CI 2-sided [-0.05 to -0.02] — Week 24. Serum Cystatin C
Statistical Analysis 2: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p = 0.022, MMRM; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.03 to 0.00] — Week 48. Serum Cystatin C
Statistical Analysis 3: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p = 0.797, MMRM; Mean Difference (Net) = -0.2, 95% CI 2-sided [-1.4 to 1.1] — Week 24. Serum RBP
Statistical Analysis 4: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p = 0.258, MMRM; Mean Difference (Net) = 0.7, 95% CI 2-sided [-0.5 to 1.9] — Week 48. Serum RBP

23. Secondary Outcome: Change From Baseline in Renal Biomarker-Serum Cystatin C at Week 96
Description: Blood and/or urine samples were collected to perform evaluation of renal biomarkers which included Serum Cystatin C. Baseline value is the latest pre-dose assessment. Change from Baseline was defined as value at indicated time point minus Baseline value. Biomarkers were adjusted for treatment, visit, Baseline plasma HIV-1 RNA, Baseline CD4+ cell count, age, sex, race, presence of diabetes mellitus, presence of hypertension, Baseline biomarker value, treatment and visit interaction, and Baseline biomarker value and visit interaction; with visit as the repeated factor. Adjusted mean and standard error is presented.
Time Frame: Baseline and at Week 96
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 316 | 326
mg/L | -0.09 (0.006) | -0.08 (0.005)
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p = 0.034, MMRM; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.03 to 0.00] — Week 96. Serum Cystatin C

24. Secondary Outcome: Change From Baseline in Renal Biomarker-Serum Cystatin C at Week 144
Description: as for outcome 23
Time Frame: Baseline and at Week 144
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 301 | 304
mg/L | -0.11 (0.005) | -0.08 (0.006)
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; p = 0.006, MMRM; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.04 to -0.01] — Week 144. Serum Cystatin C

25. Secondary Outcome: Change From Baseline in Renal Biomarker-Serum RBP at Week 96
Description: Blood and/or urine samples were collected to perform evaluation of renal biomarkers which included Serum RBP. Baseline value is the latest pre-dose assessment. Change from Baseline was defined as value at indicated time point minus Baseline value. Biomarkers were adjusted for treatment, visit, Baseline plasma HIV-1 RNA, Baseline CD4+ cell count, age, sex, race, presence of diabetes mellitus, presence of hypertension, Baseline biomarker value, treatment and visit interaction, and Baseline biomarker value and visit interaction; with visit as the repeated factor.
Time Frame: Baseline and at Week 96
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Microgram per millimoles (ug/mmol)
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 314 | 319
Microgram per millimoles (ug/mmol) | 0.557 (12.7139) | 2.483 (23.9105)

26. Secondary Outcome: Change From Baseline in Renal Biomarker-Serum RBP at Week 144
Description: as for outcome 25
Time Frame: Baseline and at Week 144
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Microgram per millimoles (ug/mmol)
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 294 | 289
Microgram per millimoles (ug/mmol) | 0.560 (9.5962) | 3.813 (10.8115)

27. Secondary Outcome: Change From Baseline in Renal Biomarkers-Serum GFR From Cystatin C Adjusted Using Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) and Serum or Plasma GFR From Creatinine Adjusted Using CKD-EPI at Weeks 24, 48
Description: Blood samples were collected to perform evaluation of renal biomarkers which included Serum GFR from cystatin C adjusted using CKD-EPI (GFR-cystatin C adjusted) and Serum or Plasma GFR from creatinine adjusted using CKD-EPI. Baseline value is the latest pre-dose Assessment. Change from Baseline was defined as value at the indicated time point minus Baseline value. Biomarkers were adjusted for treatment, visit, Baseline plasma HIV-1 RNA, baseline CD4+ cell count, age, sex, race, presence of diabetes mellitus, presence of hypertension, Baseline biomarker value, treatment and visit interaction, and Baseline biomarker value and visit interaction; with visit as the repeated factor.
Time Frame: Baseline and at Weeks 24, 48
Population: as for outcome 22
Measure: Mean (Standard Error); unit: Milliliter/minute/1.73 meter^2
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 360 | 359
Milliliter/minute/1.73 meter^2
  GFR Cystatin C adjusted, Week 24, n=345,345: number analyzed (Participants) | 345 | 345
  GFR Cystatin C adjusted, Week 24, n=345,345 | 3.8 (0.66) | 0.2 (0.65)
  GFR Cystatin C adjusted, Week 48, n=335,336: number analyzed (Participants) | 335 | 336
  GFR Cystatin C adjusted, Week 48, n=335,336 | 5.4 (0.64) | 3.6 (0.64)
  GFR creatinine adjusted, Week 24, n=346,344: number analyzed (Participants) | 346 | 344
  GFR creatinine adjusted, Week 24, n=346,344 | -12.0 (0.64) | -15.4 (0.59)
  GFR creatinine adjusted, Week 48, n=335, 337: number analyzed (Participants) | 335 | 337
  GFR creatinine adjusted, Week 48, n=335, 337 | -12.1 (0.60) | -15.4 (0.61)
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p < 0.001, MMRM; Mean Difference (Net) = 3.6, 95% CI 2-sided [1.8 to 5.4] — Week 24. GFR Cystatin C adjusted
Statistical Analysis 2: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p = 0.056, MMRM; Mean Difference (Net) = 1.7, 95% CI 2-sided [0.0 to 3.5] — Week 48. GFR Cystatin C adjusted
Statistical Analysis 3: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p < 0.001, MMRM; Mean Difference (Net) = 3.4, 95% CI 2-sided [1.7 to 5.2] — Week 24. GFR creatinine adjusted
Statistical Analysis 4: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p < 0.001, MMRM; Mean Difference (Net) = 3.3, 95% CI 2-sided [1.6 to 5.0] — Week 48. GFR creatinine adjusted

28. Secondary Outcome: Change From Baseline in Renal Biomarkers-Serum GFR From Cystatin C Adjusted Using CKD-EPI and Serum or Plasma GFR From Creatinine Adjusted for BSA Using CKD-EPI Method at Week 96
Description: Blood samples were collected to perform evaluation of renal biomarkers which included Serum GFR from cystatin C adjusted using CKD-EPI and Serum or Plasma GFR from creatinine adjusted for BSA using CKD-EPI. Baseline value is the latest pre-dose Assessment. Change from Baseline was defined as value at the indicated time point minus Baseline value. Biomarkers were adjusted for treatment, visit, Baseline plasma HIV-1 RNA, baseline CD4+ cell count, age, sex, race, presence of diabetes mellitus, presence of hypertension, Baseline biomarker value, treatment and visit interaction, and Baseline biomarker value and visit interaction; with visit as the repeated factor.
Time Frame: Baseline and at Week 96
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Milliliter/minute/1.73 meter^2
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 360 | 359
Milliliter/minute/1.73 meter^2
  GFR Cystatin C adjusted, Week 96, n=316,326: number analyzed (Participants) | 316 | 326
  GFR Cystatin C adjusted, Week 96, n=316,326 | 9.1 (18.75) | 9.5 (13.95)
  GFR creatinine adjusted, Week 96, n=315,325: number analyzed (Participants) | 315 | 325
  GFR creatinine adjusted, Week 96, n=315,325 | -14.2 (12.69) | -17.5 (11.57)

29. Secondary Outcome: Change From Baseline in Renal Biomarkers-Serum GFR From Cystatin C Adjusted Using CKD-EPI and Serum or Plasma GFR From Creatinine Adjusted for BSA Using CKD-EPI Method at Week 144
Description: as for outcome 28
Time Frame: Baseline and at Week 144
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Milliliter/minute/1.73 meter^2
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 360 | 359
Milliliter/minute/1.73 meter^2
  GFR Cystatin C adjusted, Week 144, n=301,304: number analyzed (Participants) | 301 | 304
  GFR Cystatin C adjusted, Week 144, n=301,304 | 10.3 (18.82) | 10.1 (15.50)
  GFR creatinine adjusted, Week 144, n=292,292: number analyzed (Participants) | 292 | 292
  GFR creatinine adjusted, Week 144, n=292,292 | -15.5 (12.56) | -18.2 (11.73)

30. Secondary Outcome: Change From Baseline in Renal Biomarker-Serum or Plasma Creatinine at Weeks 24, 48
Description: Blood and samples were collected to perform evaluation of renal biomarker which included Serum or Plasma Creatinine. Baseline value is defined as the the latest pre-dose assessment. Change from Baseline was calculated as value at the inidcated time point minus Baseline value. Biomarkers were adjusted for treatment, visit, Baseline plasma HIV-1 RNA, baseline CD4+ cell count, age, sex, race, presence of diabetes mellitus, presence of hypertension, Baseline biomarker value, treatment and visit interaction, and Baseline biomarker value and visit interaction; with visit as the repeated factor.
Time Frame: Baseline and at Weeks 24, 48
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Micromoles per Liter (umol/L)
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 360 | 359
Micromoles per Liter (umol/L)
  Serum or Plasma Creatinine, Week 24, n=346, 344: number analyzed (Participants) | 346 | 344
  Serum or Plasma Creatinine, Week 24, n=346, 344 | 10.51 (0.548) | 13.53 (0.507)
  Serum or Plasma Creatinine, Week 48, n=335, 337: number analyzed (Participants) | 335 | 337
  Serum or Plasma Creatinine, Week 48, n=335, 337 | 10.32 (0.519) | 13.44 (0.540)
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p < 0.001, MMRM; Mean Difference (Net) = -3.02, 95% CI 2-sided [-4.49 to -1.55] — Week 24. Serum or Plasma Creatinine
Statistical Analysis 2: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p < 0.001, MMRM; Mean Difference (Net) = -3.12, 95% CI 2-sided [-4.59 to -1.65] — Week 48. Serum or Plasma creatinine

31. Secondary Outcome: Change From Baseline in Renal Biomarker-Serum or Plasma Creatinine at Week 96
Description: Blood and samples were collected to perform evaluation of renal biomarker which included Serum or Plasma Creatinine. Baseline value is defined as the the latest pre-dose assessment. Change from Baseline was calculated as value at the inidcated time point minus Baseline value. Biomarkers were adjusted for treatment, visit, Baseline plasma HIV-1 RNA, baseline CD4+ cell count, age, sex, race, presence of diabetes mellitus, presence of hypertension, Baseline biomarker value, treatment and visit interaction, and Baseline biomarker value and visit interaction; with visit as the repeated factor. Adjusted mean and standard error has been presented.
Time Frame: Baseline and at Week 96
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Micromoles per Liter (umol/L)
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 315 | 325
Micromoles per Liter (umol/L) | 11.71 (0.563) | 14.75 (0.526)
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p < 0.001, MMRM; Mean Difference (Net) = -3.04, 95% CI 2-sided [-4.56 to -1.53] — Week 96. Serum or Plasma creatinine

32. Secondary Outcome: Change From Baseline in Renal Biomarker-Serum or Plasma Creatinine at Week 144
Description: as for outcome 31
Time Frame: Baseline and at Week 144
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Micromoles per Liter (umol/L)
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 292 | 292
Micromoles per Liter (umol/L) | 12.28 (0.613) | 15.14 (0.583)
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; p < 0.001, MMRM; Mean Difference (Net) = -2.86, 95% CI 2-sided [-4.52 to -1.19] — Week 144. Serum or Plasma creatinine

33. Secondary Outcome: Ratio to Baseline in Renal Biomarkers-Urine and Serum Beta-2 Microglobulin (B2M), Urine Albumin/Creatinine, Urine B2M/Urine Creatinine, Urine Phosphate, Urine Protein/Creatinine, Urine RBP 4 and Urine RBP 4/Urine Creatinine at Weeks 24, 48
Description: Blood and/or urine were collected to perform evaluation of renal inflammation biomarkers: Urine and Serum B2M, Urine Albumin/Creatinine, Urine B2M/Urine Creatinine, Urine Phosphate, Urine Protein/Creatinine, Urine RBP 4 and Urine RBP 4/Urine Creatinine. Baseline value was the latest pre-dose assessment. Change from Baseline was performed on log-transformed data. Ratio to Baseline was calculated as ratio of post-dose visit value over Baseline value. Geometric mean ratio and 95% CI of geometric mean ratio have been presented. Biomarkers were Adjusted for treatment, Baseline plasma HIV-1 RNA, Baseline CD4+ cell count, age, sex, race, presence of diabetes mellitus, presence of hypertension, loge transformed Baseline biomarker value, treatment and visit interaction, and loge transformed Baseline biomarker value and visit interaction; with visit as the repeated factor.
Time Frame: Baseline and Weeks 24, 48
Population: as for outcome 22
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 360 | 359
Ratio
  Serum B2M, Week 24, n=344,346: number analyzed (Participants) | 344 | 346
  Serum B2M, Week 24, n=344,346 | 0.809 [0.794 to 0.824] | 0.882 [0.867 to 0.898]
  Serum B2M, Week 48, n=335,336: number analyzed (Participants) | 335 | 336
  Serum B2M, Week 48, n=335,336 | 0.811 [0.796 to 0.827] | 0.887 [0.871 to 0.904]
  Urine B2M, Week 24, n=124,106: number analyzed (Participants) | 124 | 106
  Urine B2M, Week 24, n=124,106 | 0.844 [0.755 to 0.944] | 1.129 [0.974 to 1.309]
  Urine B2M, Week 48, n=109, 103: number analyzed (Participants) | 109 | 103
  Urine B2M, Week 48, n=109, 103 | 0.917 [0.804 to 1.046] | 1.323 [1.066 to 1.642]
  Urine Albumin/Creatinine, Week 24, n=259, 251: number analyzed (Participants) | 259 | 251
  Urine Albumin/Creatinine, Week 24, n=259, 251 | 0.907 [0.844 to 0.976] | 1.021 [0.940 to 1.109]
  Urine Albumin/Creatinine , Week 48, n=249, 240: number analyzed (Participants) | 249 | 240
  Urine Albumin/Creatinine , Week 48, n=249, 240 | 0.911 [0.835 to 0.994] | 0.971 [0.891 to 1.058]
  Urine B2M/Urine Creatinine , Week 24, n=122, 104: number analyzed (Participants) | 122 | 104
  Urine B2M/Urine Creatinine , Week 24, n=122, 104 | 0.880 [0.779 to 0.993] | 1.126 [0.988 to 1.282]
  Urine B2M/Urine Creatinine , Week 48, n=108, 103: number analyzed (Participants) | 108 | 103
  Urine B2M/Urine Creatinine , Week 48, n=108, 103 | 0.969 [0.854 to 1.099] | 1.307 [1.077 to 1.586]
  Urine Phosphate, Week 24, n=343, 340: number analyzed (Participants) | 343 | 340
  Urine Phosphate, Week 24, n=343, 340 | 1.041 [0.955 to 1.134] | 1.063 [0.978 to 1.157]
  Urine Phosphate, Week 48, n=335, 332: number analyzed (Participants) | 335 | 332
  Urine Phosphate, Week 48, n=335, 332 | 1.121 [1.031 to 1.220] | 1.056 [0.974 to 1.144]
  Urine Protein/Creatinine, Week 24, n=263,279: number analyzed (Participants) | 263 | 279
  Urine Protein/Creatinine, Week 24, n=263,279 | 0.818 [0.779 to 0.859] | 0.991 [0.941 to 1.043]
  Urine Protein/Creatinine , Week 48, n=259, 261: number analyzed (Participants) | 259 | 261
  Urine Protein/Creatinine , Week 48, n=259, 261 | 0.866 [0.818 to 0.917] | 1.007 [0.954 to 1.062]
  Urine RBP 4, Week 24, n=340, 338: number analyzed (Participants) | 340 | 338
  Urine RBP 4, Week 24, n=340, 338 | 0.656 [0.591 to 0.729] | 0.824 [0.738 to 0.921]
  Urine RBP 4, Week 48, n=333, 331: number analyzed (Participants) | 333 | 331
  Urine RBP 4, Week 48, n=333, 331 | 0.740 [0.666 to 0.822] | 0.819 [0.730 to 0.919]
  Urine RBP 4/Urine Creatinine, Week 24, n=338, 335: number analyzed (Participants) | 338 | 335
  Urine RBP 4/Urine Creatinine, Week 24, n=338, 335 | 0.670 [0.614 to 0.730] | 0.811 [0.741 to 0.888]
  Urine RBP 4/Urine Creatinine, Week 48, n=331, 328: number analyzed (Participants) | 331 | 328
  Urine RBP 4/Urine Creatinine, Week 48, n=331, 328 | 0.749 [0.689 to 0.814] | 0.844 [0.774 to 0.920]
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p < 0.001, MMRM; Ratio of geometric means = 0.917, 95% CI 2-sided [0.893 to 0.941] — Week 24. Serum B2M
Statistical Analysis 2: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p < 0.001, MMRM; Ratio of geometric means = 0.914, 95% CI 2-sided [0.890 to 0.939] — Week 48. Serum B2M
Statistical Analysis 3: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p = 0.002, MMRM; Ratio of geometric means = 0.748, 95% CI 2-sided [0.621 to 0.901] — Week 24. Urine B2M
Statistical Analysis 4: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p = 0.005, MMRM; Ratio of geometric means = 0.693, 95% CI 2-sided [0.538 to 0.892] — Week 48. Urine B2M
Statistical Analysis 5: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p = 0.036, MMRM; Ratio of geometric means = 0.889, 95% CI 2-sided [0.796 to 0.992] — Week 24. Urine Albumin/Creatinine
Statistical Analysis 6: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p = 0.308, MMRM; Ratio of geometric means = 0.938, 95% CI 2-sided [0.830 to 1.061] — Week 48. Urine Albumin/Creatinine
Statistical Analysis 7: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p = 0.007, MMRM; Ratio of geometric means = 0.781, 95% CI 2-sided [0.654 to 0.934] — Week 24. Urine B2M/Urine Creatinine
Statistical Analysis 8: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p = 0.012, MMRM; Ratio of geometric means = 0.742, 95% CI 2-sided [0.588 to 0.935] — Week 48. Urine B2M/Urine Creatinine
Statistical Analysis 9: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p = 0.728, MMRM; Ratio of geometric means = 0.979, 95% CI 2-sided [0.868 to 1.104] — Week 24. Urine Phosphate
Statistical Analysis 10: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p = 0.311, MMRM; Ratio of geometric means = 1.062, 95% CI 2-sided [0.945 to 1.194] — Week 48. Urine Phosphate
Statistical Analysis 11: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p < 0.001, MMRM; Ratio of geometric means = 0.826, 95% CI 2-sided [0.769 to 0.887] — Week 24. Urine Protein/Creatinine
Statistical Analysis 12: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p < 0.001, MMRM; Ratio of geometric means = 0.860, 95% CI 2-sided [0.795 to 0.930] — Week 48. Urine Protein/Creatinine
Statistical Analysis 13: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p = 0.003, MMRM; Ratio of geometric means = 0.796, 95% CI 2-sided [0.683 to 0.927] — Week 24. Urine RBP 4
Statistical Analysis 14: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p = 0.200, MMRM; Ratio of geometric means = 0.903, 95% CI 2-sided [0.773 to 1.056] — Week 48. Urine RBP 4
Statistical Analysis 15: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p = 0.003, MMRM; Ratio of geometric means = 0.826, 95% CI 2-sided [0.728 to 0.936] — Week 24. Urine RBP 4/Urine Creatinine
Statistical Analysis 16: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p = 0.052, MMRM; Ratio of geometric means = 0.888, 95% CI 2-sided [0.787 to 1.001] — Week 48. Urine RBP 4/Urine Creatinine

34. Secondary Outcome: Ratio to Baseline in Renal Biomarkers- Urine Albumin/Creatinine, Urine B2M/Urine Creatinine, Urine Phosphate, Urine Protein/Creatinine and Urine RBP 4/Urine Creatinine at Week 96
Description: Blood and/or urine were collected to perform evaluation of renal inflammation biomarkers: Urine Albumin/Creatinine, Urine B2M/Urine Creatinine, Urine Phosphate, Urine Protein/Creatinine and Urine RBP 4/Urine Creatinine. Baseline value was the latest pre-dose assessment. Change from Baseline was performed on log-transformed data. Ratio to Baseline was calculated as ratio of post-dose visit value over Baseline value. Biomarkers were Adjusted for treatment, Baseline plasma HIV-1 RNA, Baseline CD4+ cell count, age, sex, race, presence of diabetes mellitus, presence of hypertension, loge transformed Baseline biomarker value, treatment and visit interaction, and loge transformed Baseline biomarker value and visit interaction; with visit as the repeated factor.
Time Frame: Baseline and Week 96
Population: as for outcome 22
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 360 | 359
Ratio
  Urine Albumin/Creatinine, Week 96, n=239, 243: number analyzed (Participants) | 239 | 243
  Urine Albumin/Creatinine, Week 96, n=239, 243 | 0.939 [0.861 to 1.023] | 0.997 [0.914 to 1.087]
  Urine B2M/Urine Creatinine, Week 96, n=101, 96: number analyzed (Participants) | 101 | 96
  Urine B2M/Urine Creatinine, Week 96, n=101, 96 | 0.844 [0.757 to 0.941] | 1.259 [1.055 to 1.503]
  Urine Phosphate, Week 96, n=316, 322: number analyzed (Participants) | 316 | 322
  Urine Phosphate, Week 96, n=316, 322 | 1.156 [1.064 to 1.256] | 1.069 [0.988 to 1.156]
  Urine Protein/Creatinine, Week 96, n=251, 261: number analyzed (Participants) | 251 | 261
  Urine Protein/Creatinine, Week 96, n=251, 261 | 0.887 [0.836 to 0.942] | 1.016 [0.963 to 1.072]
  Urine RBP 4/Urine Creatinine, Week 96, n=314, 318: number analyzed (Participants) | 314 | 318
  Urine RBP 4/Urine Creatinine, Week 96, n=314, 318 | 1.030 [0.953 to 1.113] | 1.287 [1.189 to 1.393]
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p = 0.338, MMRM; Ratio of geometric means = 0.942, 95% CI 2-sided [0.833 to 1.065] — Week 96. Urine Albumin/Creatinine
Statistical Analysis 2: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p < 0.001, MMRM; Ratio of geometric means = 0.671, 95% CI 2-sided [0.545 to 0.826] — Week 96. Urine B2M/Urine Creatinine
Statistical Analysis 3: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p = 0.174, MMRM; Ratio of geometric means = 1.082, 95% CI 2-sided [0.966 to 1.213] — Week 96. Urine Phosphate
Statistical Analysis 4: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p < 0.001, MMRM; Ratio of geometric means = 0.873, 95% CI 2-sided [0.806 to 0.946] — Week 96. Urine Protein/Creatinine
Statistical Analysis 5: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p < 0.001, MMRM; Ratio of geometric means = 0.800, 95% CI 2-sided [0.716 to 0.894] — Week 96. Urine RBP 4/Urine Creatinine

35. Secondary Outcome: Ratio to Baseline in Renal Biomarkers- Urine Albumin/Creatinine, Urine B2M/Urine Creatinine, Urine Phosphate, Urine Protein/Creatinine and Urine RBP 4/Urine Creatinine at Week 144
Description: as for outcome 34
Time Frame: Baseline and at Week 144
Population: as for outcome 22
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 360 | 359
Ratio
  Urine Albumin/Creatinine, Week 144, n=230, 221: number analyzed (Participants) | 230 | 221
  Urine Albumin/Creatinine, Week 144, n=230, 221 | 1.036 [0.943 to 1.138] | 1.067 [0.973 to 1.169]
  Urine B2M/Urine Creatinine, Week 144, n=108, 93: number analyzed (Participants) | 108 | 93
  Urine B2M/Urine Creatinine, Week 144, n=108, 93 | 0.872 [0.792 to 0.960] | 1.494 [1.266 to 1.762]
  Urine Phosphate, Week 144, n=301, 301: number analyzed (Participants) | 301 | 301
  Urine Phosphate, Week 144, n=301, 301 | 1.083 [1.000 to 1.174] | 1.084 [0.999 to 1.175]
  Urine Protein/Creatinine, Week 144, n=236, 246: number analyzed (Participants) | 236 | 246
  Urine Protein/Creatinine, Week 144, n=236, 246 | 0.999 [0.947 to 1.054] | 1.180 [1.118 to 1.245]
  Urine RBP 4/Urine Creatinine, Week 144, n=294, 289: number analyzed (Participants) | 294 | 289
  Urine RBP 4/Urine Creatinine, Week 144, n=294, 289 | 1.159 [1.083 to 1.240] | 1.567 [1.451 to 1.694]
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; p = 0.658, MMRM; Ratio of geometric means = 0.971, 95% CI 2-sided [0.852 to 1.107] — Week 144. Urine Albumin/Creatinine
Statistical Analysis 2: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; p < 0.001, MMRM; Ratio of geometric means = 0.584, 95% CI 2-sided [0.483 to 0.706] — Week 144. Urine B2M/Urine Creatinine
Statistical Analysis 3: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; p = 0.993, MMRM; Ratio of geometric means = 1.000, 95% CI 2-sided [0.892 to 1.120] — Week 144. Urine Phosphate
Statistical Analysis 4: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; p < 0.001, MMRM; Ratio of geometric means = 0.847, 95% CI 2-sided [0.785 to 0.913] — Week 144. Urine Protein/Creatinine
Statistical Analysis 5: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; p < 0.001, MMRM; Ratio of geometric means = 0.739, 95% CI 2-sided [0.667 to 0.819] — Week 144. Urine RBP 4/Urine Creatinine

36. Secondary Outcome: Change From Baseline in Bone Biomarkers-Serum Bone Specific Alkaline Phosphatase (Bone-ALP), Serum Osteocalcin, Serum Procollagen 1 N-Terminal Propeptide (PINP) and Serum Type I Collagen C-Telopeptides (CTX-1) at Weeks 24, 48
Description: Blood samples were collected to perform evaluation of bone biomarkers which included bone-ALP, Serum Osteocalcin, PINP and CTX-1. Adjusted mean and standard error is presented. Adjusted mean is the estimated mean change from Baseline at each visit in each arm calculated from a repeated measures model adjusting for: treatment, visit, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count (factor), age, sex (factor), race (factor), BMI (factor), smoking status (factor), current Vitamin D use (factor), Baseline biomarker value, treatment and visit interaction, and Baseline biomarker value and visit interaction; with visit as the repeated factor. Baseline value is defined as the latest pre-dose assessment. Change from Baseline was calculated as value at the indicated time point minus Baseline value.
Time Frame: Baseline (Day 1) and at Weeks 24, 48
Population: as for outcome 22
Measure: Mean (Standard Error); unit: Micrograms per Liter (ug/L)
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 360 | 359
Micrograms per Liter (ug/L)
  Bone-ALP, Week 24, n=345, 346: number analyzed (Participants) | 345 | 346
  Bone-ALP, Week 24, n=345, 346 | 0.72 (0.171) | 3.38 (0.244)
  Bone-ALP, Week 48, n=334, 337: number analyzed (Participants) | 334 | 337
  Bone-ALP, Week 48, n=334, 337 | 1.24 (0.198) | 4.33 (0.268)
  Serum Osteocalcin, Week 24, n=345, 346: number analyzed (Participants) | 345 | 346
  Serum Osteocalcin, Week 24, n=345, 346 | 2.13 (0.321) | 6.80 (0.368)
  Serum Osteocalcin, Week 48, n=335, 336: number analyzed (Participants) | 335 | 336
  Serum Osteocalcin, Week 48, n=335, 336 | 0.40 (0.326) | 6.30 (0.384)
  PINP, Week 24, n=344, 346: number analyzed (Participants) | 344 | 346
  PINP, Week 24, n=344, 346 | 1.7 (0.95) | 15.2 (1.12)
  PINP, Week 48, n=335, 337: number analyzed (Participants) | 335 | 337
  PINP, Week 48, n=335, 337 | 0.4 (0.79) | 13.3 (1.06)
  CTX-1, Week 24, n=342, 342: number analyzed (Participants) | 342 | 342
  CTX-1, Week 24, n=342, 342 | 0.1541 (0.01247) | 0.2812 (0.01406)
  CTX-1, Week 48, n=332, 333: number analyzed (Participants) | 332 | 333
  CTX-1, Week 48, n=332, 333 | 0.1345 (0.01496) | 0.3388 (0.01983)
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p < 0.001, MMRM; Mean Difference (Net) = -2.66, 95% CI 2-sided [-3.25 to -2.08] — Week 24, Bone ALP
Statistical Analysis 2: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p < 0.001, MMRM; Mean Difference (Net) = -3.09, 95% CI 2-sided [-3.75 to -2.44] — Week 48, Bone ALP
Statistical Analysis 3: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p < 0.001, MMRM; Mean Difference (Net) = -4.67, 95% CI 2-sided [-5.63 to -3.71] — Week 28, Serum Osteocalcin
Statistical Analysis 4: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p < 0.001, MMRM; Mean Difference (Net) = -5.90, 95% CI 2-sided [-6.89 to -4.91] — Week 48, Serum Osteocalcin
Statistical Analysis 5: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p < 0.001, MMRM; Mean Difference (Net) = -13.5, 95% CI 2-sided [-16.4 to -10.6] — Week 24, Serum PINP
Statistical Analysis 6: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p < 0.001, MMRM; Mean Difference (Net) = -12.8, 95% CI 2-sided [-15.4 to -10.2] — Week 48, Serum PINP
Statistical Analysis 7: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p < 0.001, MMRM; Mean Difference (Net) = -0.1270, 95% CI 2-sided [-0.1640 to -0.0900] — Week 24, CTX-1
Statistical Analysis 8: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p < 0.001, MMRM; Mean Difference (Net) = -0.2043, 95% CI 2-sided [-0.2532 to -0.1554] — Week 48, CTX-1

37. Secondary Outcome: Change From Baseline in Bone Biomarkers-Serum Bone-ALP, Serum Osteocalcin, Serum PINP and Serum Type I CTX-1 at Week 96
Description: Blood samples were collected to perform evaluation of bone biomarkers which included bone-ALP, Serum Osteocalcin, Serum PINP and Serum Type CTX-1. Adjusted mean is the estimated mean change from Baseline in each arm calculated from a repeated measures model adjusting for: treatment, visit, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count (factor), age, sex (factor), race (factor), BMI (factor), smoking status (factor), current vitamin D use (factor), Baseline biomarker value, treatment and visit interaction, and Baseline biomarker value and visit interaction; with visit as the repeated factor. Baseline value is defined as the latest pre-dose assessment. Change from Baseline was calculated as value at the indicated time point minus Baseline value. Adjusted mean and standard error is presented.
Time Frame: Baseline (Day 1) and at Week 96
Population: as for outcome 22
Measure: Mean (Standard Error); unit: Micrograms per Liter (ug/L)
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 360 | 359
Micrograms per Liter (ug/L)
  Bone-ALP, Week 96, n=315, 326: number analyzed (Participants) | 315 | 326
  Bone-ALP, Week 96, n=315, 326 | 0.26 (0.188) | 2.39 (0.234)
  Serum Osteocalcin, Week 96, n=315, 326: number analyzed (Participants) | 315 | 326
  Serum Osteocalcin, Week 96, n=315, 326 | 0.13 (0.286) | 3.90 (0.368)
  PINP, Week 96, n=315, 325: number analyzed (Participants) | 315 | 325
  PINP, Week 96, n=315, 325 | 7.0 (1.37) | 19.5 (1.66)
  CTX-1, Week 96, n=311, 318: number analyzed (Participants) | 311 | 318
  CTX-1, Week 96, n=311, 318 | 0.0604 (0.01056) | 0.1787 (0.01403)
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p < 0.001, MMRM; Mean Difference (Net) = -2.13, 95% CI 2-sided [-2.72 to -1.54] — Week 96, Bone ALP
Statistical Analysis 2: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p < 0.001, MMRM; Mean Difference (Net) = -3.77, 95% CI 2-sided [-4.69 to -2.85] — Week 96, Serum Osteocalcin
Statistical Analysis 3: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p < 0.001, MMRM; Mean Difference (Net) = -12.6, 95% CI 2-sided [-16.8 to -8.3] — Week 96, Serum PINP
Statistical Analysis 4: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p < 0.001, MMRM; Mean Difference (Net) = -0.1183, 95% CI 2-sided [-0.1529 to -0.0838] — Week 96, CTX-1

38. Secondary Outcome: Change From Baseline in Bone Biomarkers-Serum Bone-ALP, Serum Osteocalcin, Serum PINP and Serum Type I CTX-1 at Week 144
Description: as for outcome 37
Time Frame: Baseline (Day 1) and at Week 144
Population: as for outcome 22
Measure: Mean (Standard Error); unit: Micrograms per Liter (ug/L)
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 360 | 359
Micrograms per Liter (ug/L)
  Bone-ALP, Week 144, n=302, 305: number analyzed (Participants) | 302 | 305
  Bone-ALP, Week 144, n=302, 305 | -0.25 (0.156) | 1.88 (0.266)
  Serum Osteocalcin, Week 144, n=300, 304: number analyzed (Participants) | 300 | 304
  Serum Osteocalcin, Week 144, n=300, 304 | -1.02 (0.280) | 2.87 (0.412)
  PINP, Week 144, n=299, 300: number analyzed (Participants) | 299 | 300
  PINP, Week 144, n=299, 300 | -0.1 (0.94) | 9.4 (1.39)
  CTX-1, Week 144, n=291, 298: number analyzed (Participants) | 291 | 298
  CTX-1, Week 144, n=291, 298 | 0.0505 (0.01154) | 0.1868 (0.01516)
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; p < 0.001, MMRM; Mean Difference (Net) = -2.13, 95% CI 2-sided [-2.74 to -1.53] — Week 144, Bone ALP
Statistical Analysis 2: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; p < 0.001, MMRM; Mean Difference (Net) = -3.89, 95% CI 2-sided [-4.87 to -2.91] — Week 144, Serum Osteocalcin
Statistical Analysis 3: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; p < 0.001, MMRM; Mean Difference (Net) = -9.5, 95% CI 2-sided [-12.8 to -6.2] — Week 144, Serum PINP
Statistical Analysis 4: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; p < 0.001, MMRM; Mean Difference (Net) = -0.1364, 95% CI 2-sided [-0.1739 to -0.0988] — Week 144, CTX-1

39. Secondary Outcome: Change From Baseline in Bone Biomarker-Serum Vitamin D at Weeks 24, 48
Description: Blood samples were collected to perform evaluation of bone biomarker serum vitamin D. Adjusted mean and standard error is presented. Adjusted mean is the estimated mean change from Baseline at each visit in each arm calculated from a repeated measures model adjusting for: treatment, visit, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count (factor), age, sex (factor), race (factor), BMI (factor), smoking status (factor), current Vitamin D use (factor), Baseline biomarker value, treatment and visit interaction, and Baseline biomarker value and visit interaction; with visit as the repeated factor. Baseline value is defined as the latest pre-dose assessment. Change from Baseline was calculated as value at the indicated time point minus Baseline value.
Time Frame: Baseline and at Weeks 24, 48
Population: as for outcome 22
Measure: Least Squares Mean (Standard Error); unit: Nanomoles per Liter (nmol/L)
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 360 | 359
Nanomoles per Liter (nmol/L)
  Serum Vitamin D, Week 24, n=346, 344: number analyzed (Participants) | 346 | 344
  Serum Vitamin D, Week 24, n=346, 344 | 11.2 (1.08) | 15.4 (1.33)
  Serum Vitamin D, Week 48, n=336, 335: number analyzed (Participants) | 336 | 335
  Serum Vitamin D, Week 48, n=336, 335 | 0.3 (0.92) | 0.4 (1.01)
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p = 0.015, MMRM; Mean Difference (Net) = -4.2, 95% CI 2-sided [-7.5 to -0.8] — Week 24
Statistical Analysis 2: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p = 0.960, MMRM; Mean Difference (Net) = -0.1, 95% CI 2-sided [-2.8 to 2.6] — Week 48

40. Secondary Outcome: Change From Baseline in Bone Biomarker-Serum Vitamin D at Week 96
Description: as for outcome 39
Time Frame: Baseline and at Week 96
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Nanomoles per Liter (nmol/L)
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 312 | 326
Nanomoles per Liter (nmol/L) | -1.7 (1.01) | 1.3 (1.09)
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p = 0.048, MMRM; Mean Difference (Net) = -3.0, 95% CI 2-sided [-5.9 to 0.0] — Week 96, Serum Vitamin D

41. Secondary Outcome: Change From Baseline in Bone Biomarker-Serum Vitamin D at Week 144
Description: as for outcome 39
Time Frame: Baseline and at Week 144
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Nanomoles per Liter (nmol/L)
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 303 | 303
Nanomoles per Liter (nmol/L) | 1.1 (1.20) | 1.4 (1.22)
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; p = 0.887, MMRM; Mean Difference (Net) = -0.2, 95% CI 2-sided [-3.6 to 3.1] — Week 144, Serum Vitamin D

42. Secondary Outcome: Percentage Change From Baseline in Fasting Lipids-Serum or Plasma Cholesterol, Serum or Plasma High Density Lipoprotein (HDL) Cholesterol (Direct), Serum or Plasma LDL Cholesterol (Calculated or Direct) and Serum or Plasma Triglycerides at Weeks 24, 48
Description: Blood samples were collected to perform evaluation of fasting lipids which included Serum or Plasma Cholesterol, Serum or Plasma HDL Cholesterol (Direct), Serum or Plasma LDL Cholesterol (Calculated or Direct) and Serum or Plasma Triglycerides. Baseline value is defined as the latest pre-dose assessment (Day 1). Percentage change from Baseline was calculated as 100 multiplied by ([post-dose visit value minus Baseline value] divided by Baseline value).
Time Frame: Baseline and at Weeks 24, 48
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 360 | 359
Percentage change
  Serum or Plasma Cholesterol, Week 24, n=298, 310: number analyzed (Participants) | 298 | 310
  Serum or Plasma Cholesterol, Week 24, n=298, 310 | 5.0 (16.85) | -4.5 (15.44)
  Serum or Plasma Cholesterol, Week 48, n=298, 307: number analyzed (Participants) | 298 | 307
  Serum or Plasma Cholesterol, Week 48, n=298, 307 | 9.3 (17.10) | -3.3 (14.61)
  HDL Cholesterol, Direct, Week 24, n=299, 310: number analyzed (Participants) | 299 | 310
  HDL Cholesterol, Direct, Week 24, n=299, 310 | 13.9 (25.17) | 7.2 (32.22)
  HDL Cholesterol, Direct, Week 48, n=299, 307: number analyzed (Participants) | 299 | 307
  HDL Cholesterol, Direct, Week 48, n=299, 307 | 15.3 (23.75) | 4.0 (21.86)
  LDL Cholesterol, Week 24, n=298, 309: number analyzed (Participants) | 298 | 309
  LDL Cholesterol, Week 24, n=298, 309 | 3.8 (25.85) | -7.8 (21.13)
  LDL Cholesterol, Week 48, n=297, 307: number analyzed (Participants) | 297 | 307
  LDL Cholesterol, Week 48, n=297, 307 | 10.7 (27.54) | -4.1 (20.39)
  Triglycerides,Week 24, n=299, 310: number analyzed (Participants) | 299 | 310
  Triglycerides,Week 24, n=299, 310 | 7.0 (40.45) | 0.5 (44.01)
  Triglycerides, Week 48, n=299, 307: number analyzed (Participants) | 299 | 307
  Triglycerides, Week 48, n=299, 307 | 7.3 (46.92) | -0.3 (49.22)

43. Secondary Outcome: Change From Baseline in Fasting Lipids-Serum or Plasma Cholesterol, Serum or Plasma HDL Cholesterol (Direct), Serum or Plasma LDL Cholesterol (Calculated or Direct) and Serum or Plasma Triglycerides at Week 96
Description: Blood samples were collected to perform evaluation of fasting lipids which included Serum or Plasma Cholesterol, Serum or Plasma HDL Cholesterol (Direct), Serum or Plasma LDL Cholesterol (Calculated or Direct) and Serum or Plasma Triglycerides. Baseline value was defined as the latest pre-dose assessment (Day 1). Change from Baseline was defined as value at the indicated time point minus Baseline value. Adjusted mean and standard error is presented.
Time Frame: Baseline (Day 1) and at Week 96
Population: as for outcome 22
Measure: Mean (Standard Error); unit: Millimoles per liter
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 360 | 359
Millimoles per liter
  Serum or Plasma Cholesterol, Week 96, n=270, 289: number analyzed (Participants) | 270 | 289
  Serum or Plasma Cholesterol, Week 96, n=270, 289 | 0.345 (0.0356) | -0.132 (0.0375)
  HDL Cholesterol, Direct, Week 96, n=271, 289: number analyzed (Participants) | 271 | 289
  HDL Cholesterol, Direct, Week 96, n=271, 289 | 0.185 (0.0160) | 0.071 (0.0136)
  LDL Cholesterol, Week 96, n=270, 289: number analyzed (Participants) | 270 | 289
  LDL Cholesterol, Week 96, n=270, 289 | 0.139 (0.0308) | -0.160 (0.0304)
  Triglycerides, Week 96, n=271, 289: number analyzed (Participants) | 271 | 289
  Triglycerides, Week 96, n=271, 289 | 0.105 (0.0488) | -0.102 (0.0365)

44. Secondary Outcome: Change From Baseline in Fasting Lipids-Serum or Plasma Cholesterol, Serum or Plasma HDL Cholesterol (Direct), Serum or Plasma LDL Cholesterol (Calculated or Direct) and Serum or Plasma Triglycerides at Week 144
Description: as for outcome 43
Time Frame: Baseline (Day 1) and at Week 144
Population: as for outcome 22
Measure: Mean (Standard Error); unit: Millimoles per liter
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 360 | 359
Millimoles per liter
  Serum or Plasma Cholesterol, Week 144, n=263, 278: number analyzed (Participants) | 263 | 278
  Serum or Plasma Cholesterol, Week 144, n=263, 278 | 0.360 (0.0432) | -0.015 (0.0394)
  HDL Cholesterol, Direct, Week 144, n=264, 278: number analyzed (Participants) | 264 | 278
  HDL Cholesterol, Direct, Week 144, n=264, 278 | 0.180 (0.0162) | 0.093 (0.0136)
  LDL Cholesterol, Week 144, n=263, 278: number analyzed (Participants) | 263 | 278
  LDL Cholesterol, Week 144, n=263, 278 | 0.143 (0.0357) | -0.085 (0.0333)
  Triglycerides, Week 144, n=264, 278: number analyzed (Participants) | 264 | 278
  Triglycerides, Week 144, n=264, 278 | 0.078 (0.0448) | -0.057 (0.0430)

45. Secondary Outcome: Percentage Change From Baseline in Fasting Lipid-Serum or Plasma Total Cholesterol/HDL Cholesterol Ratio at Weeks 24, 48
Description: Blood samples were collected to perform evaluation of fasting lipid-Serum or Plasma Total Cholesterol/HDL Cholesterol Ratio. Baseline value is the latest pre-dose assessment (Day 1). Percentage change from Baseline was calculated as 100 multiplied by ([post-dose visit value minus Baseline value] divided by Baseline value). Lipid last observation carried forwarded (LOCF) data was used such that the last available fasted, on-treatment lipid value prior to the initiation of a lipid-lowering agent was used in place of future observed values. Participants on lipid-lowering agents at Baseline were excluded.
Time Frame: Baseline (Day 1) and at Weeks 24, 48
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 360 | 359
Percentage change
  Total/HDL Cholesterol Ratio, Week 24, n=298, 310: number analyzed (Participants) | 298 | 310
  Total/HDL Cholesterol Ratio, Week 24, n=298, 310 | -4.4 (22.53) | -7.5 (17.90)
  Total/HDL Cholesterol Ratio, Week 48, n=298, 307: number analyzed (Participants) | 298 | 307
  Total/HDL Cholesterol Ratio, Week 48, n=298, 307 | -2.8 (17.86) | -4.5 (18.25)

46. Secondary Outcome: Change From Baseline in Fasting Lipid-Serum or Plasma Total Cholesterol/HDL Cholesterol Ratio at Week 96
Description: Blood samples were collected to perform evaluation of fasting lipid-Serum or Plasma Total Cholesterol/HDL Cholesterol Ratio. Baseline value is the latest pre-dose assessment (Day 1). Baseline value was defined as the latest pre-dose assessment (Day 1). Change from Baseline was defined as value at the indicated time point minus Baseline value. Adjusted mean and standard error is presented.
Time Frame: Baseline (Day 1) and at Week 96
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 270 | 289
Ratio | -0.113 (0.1552) | -0.395 (0.0473)

47. Secondary Outcome: Change From Baseline in Fasting Lipid-Serum or Plasma Total Cholesterol/HDL Cholesterol Ratio at Week 144
Description: as for outcome 46
Time Frame: Baseline (Day 1) and at Week 144
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 263 | 278
Ratio | -0.245 (0.0545) | -0.359 (0.0533)

48. Secondary Outcome: Percentage of Participants With Grade 2 or Greater Laboratory Abnormalities in Fasting LDL Cholesterol by Weeks 24, 48
Description: Blood samples were collected to perform evaluation of fasting LDL cholesterol. Any abnormalities were evaluated by the investigator and graded according to DAIDS toxicity scales from Grade 1 to 4 (1=Mild, 2=Moderate, 3=Severe, 4=Potentially life threatening). The higher the grade, the more severe the symptoms. Percentage of participants with Grade 2 or greater laboratory abnormalities in fasting LDL cholesterol by Weeks 24 and 48 have been presented. Participants without any post-Baseline fasting LDL cholesterol value prior to Week 48 or those who had Baseline lipids-lowering agents were not included. Lipid Last Observation Carried Forward (LOCF) data was used such that the last available fasted, on-treatment lipid value prior to the initiation of a lipid-lowering agent was used in place of future observed values. Percentage values are rounded-off.
Time Frame: Weeks 24 and 48
Population: as for outcome 22
Measure: Number; unit: Percentage of participants
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 360 | 359
Percentage of participants
  Week 24, n=313, 320: number analyzed (Participants) | 313 | 320
  Week 24, n=313, 320 | 4 | 0
  Week 48, n=324, 332: number analyzed (Participants) | 324 | 332
  Week 48, n=324, 332 | 4 | 2
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p < 0.001, Fisher Exact; Mean Difference (Final Values) = 3.5, 95% CI 2-sided [1.5 to 5.6] — Week 24
Statistical Analysis 2: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p = 0.037, Fisher Exact; Mean Difference (Final Values) = 2.8, 95% CI 2-sided [0.2 to 5.4] — Week 48

49. Secondary Outcome: Percentage of Participants With Grade 2 or Greater Laboratory Abnormalities in Fasting LDL Cholesterol by Week 96
Description: Blood samples were collected to perform evaluation of fasting LDL cholesterol. Any abnormalities were evaluated by the investigator and graded according to DAIDS toxicity scales from Grade 1 to 4 (1=Mild, 2=Moderate, 3=Severe, 4=Potentially life threatening). The higher the grade, the more severe the symptoms. Percentage of participants with Grade 2 or greater laboratory abnormalities in fasting LDL cholesterol by Week 96 have been presented. Participants without any post-Baseline fasting LDL cholesterol value prior to Week 96 or those who had Baseline lipids-lowering agents were not included. Lipid Last Observation Carried Forward (LOCF) data was used such that the last available fasted, on-treatment lipid value prior to the initiation of a lipid-lowering agent was used in place of future observed values. Percentage values are rounded-off.
Time Frame: Week 96
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 324 | 332
Percentage of participants | 6 | 2
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p = 0.045, Fisher Exact; Mean Difference (Final Values) = 3.1, 95% CI 2-sided [0.2 to 6.1] — Week 96

50. Secondary Outcome: Percentage of Participants With Grade 2 or Greater Laboratory Abnormalities in Fasting LDL Cholesterol by Week 144
Description: Blood samples were collected to perform evaluation of fasting LDL cholesterol. Any abnormalities were evaluated by the investigator and graded according to DAIDS toxicity scales from Grade 1 to 4 (1=Mild, 2=Moderate, 3=Severe, 4=Potentially life threatening). Percentage of participants with Grade 2 or greater laboratory abnormalities in fasting LDL cholesterol by Week 144 have been presented. Participants without any post-Baseline fasting LDL cholesterol value prior to Week 144 or those who had Baseline lipids-lowering agents were not included. Lipid Last Observation Carried Forward (LOCF) data was used such that the last available fasted, on-treatment lipid value prior to the initiation of a lipid-lowering agent was used in place of future observed values. Percentage values are rounded-off.
Time Frame: Week 144
Population: Safety Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 324 | 333
Percentage of participants | 6 | 4
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; p = 0.160, Fisher Exact; Mean Difference (Final Values) = 2.6, 95% CI 2-sided [-0.8 to 6.0] — Week 144

51. Secondary Outcome: Percentage of Participants by Subgroups (by Age, Gender, Baseline CD4+ Cell Count, Baseline HIV-1 RNA, Race) With Plasma HIV-1 RNA <50 c/mL at Week 24
Description: Percentage of participants by subgroups (by age, gender, Baseline CD4+ cell count, Baseline HIV-1 RNA, race) with HIV-1 RNA<50 c/mL was obtained using FDA Snapshot algorithm. The Snapshot algorithm treated all participants without HIV-1 RNA data at the visit of interest (due to missing data or discontinuation of investigational product prior to the visit window) as non-responders, as well as participants who switch their concomitant ART prior to the visit of interest. Data was presented by subgroups: age (<35, 35 to <50, >=50 years); gender (males and females), Baseline CD4+ cell count (<=200 cells/mm^3, >200 cells/mm^3 for group-1), Baseline HIV-1 RNA (<=100000, >100000 c/mL) and Race (White, African American/African heritage (H.), Asian other). Percentage values are rounded-off.
Time Frame: Week 24
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 360 | 359
Percentage of participants
  Baseline CD4+ cell count Group-1, <=200,n=32,26: number analyzed (Participants) | 32 | 26
  Baseline CD4+ cell count Group-1, <=200,n=32,26 | 78 | 92
  Baseline CD4+ cell count Group-1, >200,n=328,333: number analyzed (Participants) | 328 | 333
  Baseline CD4+ cell count Group-1, >200,n=328,333 | 95 | 94
  Female, n=54, 46: number analyzed (Participants) | 54 | 46
  Female, n=54, 46 | 93 | 89
  Male, n=306, 313: number analyzed (Participants) | 306 | 313
  Male, n=306, 313 | 94 | 95
  Age, <35,n= 209, 203: number analyzed (Participants) | 209 | 203
  Age, <35,n= 209, 203 | 93 | 94
  Age, 35 to <50,n=115, 122: number analyzed (Participants) | 115 | 122
  Age, 35 to <50,n=115, 122 | 96 | 94
  Age, >=50, n=36, 34: number analyzed (Participants) | 36 | 34
  Age, >=50, n=36, 34 | 94 | 91
  Baseline plasma HIV-1 RNA, <=100000,n=294,282: number analyzed (Participants) | 294 | 282
  Baseline plasma HIV-1 RNA, <=100000,n=294,282 | 94 | 95
  Baseline plasma HIV-1 RNA, >100000,n=66, 77: number analyzed (Participants) | 66 | 77
  Baseline plasma HIV-1 RNA, >100000,n=66, 77 | 92 | 90
  Race, White, n=240, 252: number analyzed (Participants) | 240 | 252
  Race, White, n=240, 252 | 95 | 95
  Race, African American/African H., n=51, 35: number analyzed (Participants) | 51 | 35
  Race, African American/African H., n=51, 35 | 90 | 89
  Race, Asian, n=34, 30: number analyzed (Participants) | 34 | 30
  Race, Asian, n=34, 30 | 97 | 90
  Race, Other, n=35, 42: number analyzed (Participants) | 35 | 42
  Race, Other, n=35, 42 | 89 | 93

52. Secondary Outcome: Percentage of Participants by Subgroups (by Age, Gender, Baseline CD4+ Cell Count Baseline HIV-1 RNA, Race) With Plasma HIV-1 RNA <50 c/mL at Week 48
Description: Percentage of participants by subgroups (by age, gender, Baseline CD4+ cell count, Baseline HIV-1 RNA, race) with HIV-1 RNA<50 c/mL was obtained using FDA Snapshot algorithm. The Snapshot algorithm treated all participants without HIV-1 RNA data at the visit of interest (due to missing data or discontinuation of investigational product prior to the visit window) as non-responders, as well as participants who switch their concomitant ART prior to the visit of interest. Data was presented by subgroups: age (<35, 35 to <50, >=50 years); gender (males and females), Baseline CD4+ cell count (<=200 cells/mm^3, >200 cells/mm^3 for group-1), Baseline HIV-1 RNA (<=100000, >100000) and Race (White, African American/African H., Asian and other). Percentage values are rounded-off.
Time Frame: Week 48
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 360 | 359
Percentage of participants
  Baseline CD4+ cell count Group-1, <=200,n=32, 26: number analyzed (Participants) | 32 | 26
  Baseline CD4+ cell count Group-1, <=200,n=32, 26 | 78 | 96
  Baseline CD4+ cell count Group-1, >200,n=328,333: number analyzed (Participants) | 328 | 333
  Baseline CD4+ cell count Group-1, >200,n=328,333 | 95 | 94
  Female, n=54, 46: number analyzed (Participants) | 54 | 46
  Female, n=54, 46 | 89 | 87
  Male, n=306, 313: number analyzed (Participants) | 306 | 313
  Male, n=306, 313 | 94 | 95
  Age, <35,n= 209,203: number analyzed (Participants) | 209 | 203
  Age, <35,n= 209,203 | 92 | 94
  Age, 35 to <50,n=115, 122: number analyzed (Participants) | 115 | 122
  Age, 35 to <50,n=115, 122 | 97 | 94
  Age, >=50, n=36, 34: number analyzed (Participants) | 36 | 34
  Age, >=50, n=36, 34 | 89 | 94
  Baseline plasma HIV-1 RNA, <=100000,n=294,282: number analyzed (Participants) | 294 | 282
  Baseline plasma HIV-1 RNA, <=100000,n=294,282 | 92 | 95
  Baseline plasma HIV-1 RNA, >100000,n=66, 77: number analyzed (Participants) | 66 | 77
  Baseline plasma HIV-1 RNA, >100000,n=66, 77 | 97 | 90
  Race, White, n=240, 252: number analyzed (Participants) | 240 | 252
  Race, White, n=240, 252 | 96 | 96
  Race, African American/African H., n=51, 35: number analyzed (Participants) | 51 | 35
  Race, African American/African H., n=51, 35 | 80 | 86
  Race, Asian, n=34, 30: number analyzed (Participants) | 34 | 30
  Race, Asian, n=34, 30 | 97 | 90
  Race, Other, n=35, 42: number analyzed (Participants) | 35 | 42
  Race, Other, n=35, 42 | 86 | 90

53. Secondary Outcome: Percentage of Participants by Subgroups (by Age, Gender, Baseline CD4+ Cell Count Baseline HIV-1 RNA, Race) With Plasma HIV-1 RNA <50 c/mL at Week 96
Description: Percentage of participants by subgroups (by age, gender, Baseline CD4+ cell count, Baseline HIV-1 RNA, race) with HIV-1 RNA<50 c/mL was obtained using FDA Snapshot algorithm. The Snapshot algorithm treated all participants without HIV-1 RNA data at the visit of interest (due to missing data or discontinuation of investigational product prior to the visit window) as non-responders, as well as participants who switch their concomitant ART prior to the visit of interest. Data was presented by subgroups: age (<35, 35 to <50, >=50 years); gender (males and females), Baseline CD4+ cell count (<=200 cells/mm^3, >200 cells/mm^3), Baseline HIV-1 RNA (<=100000, >100000) and Race (White, African American/African H., Asian and other). Percentage values are rounded-off.
Time Frame: Week 96
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 360 | 359
Percentage of participants
  Baseline CD4+ cell count, <=200,n=32, 26: number analyzed (Participants) | 32 | 26
  Baseline CD4+ cell count, <=200,n=32, 26 | 72 | 85
  Baseline CD4+ cell count, >200,n=328,333: number analyzed (Participants) | 328 | 333
  Baseline CD4+ cell count, >200,n=328,333 | 89 | 90
  Female, n=54, 46: number analyzed (Participants) | 54 | 46
  Female, n=54, 46 | 81 | 85
  Male, n=306, 313: number analyzed (Participants) | 306 | 313
  Male, n=306, 313 | 89 | 90
  Age, <35,n= 209, 203: number analyzed (Participants) | 209 | 203
  Age, <35,n= 209, 203 | 88 | 91
  Age, 35 to <50,n=115, 122: number analyzed (Participants) | 115 | 122
  Age, 35 to <50,n=115, 122 | 90 | 89
  Age, >=50, n=36, 34: number analyzed (Participants) | 36 | 34
  Age, >=50, n=36, 34 | 83 | 88
  Baseline plasma HIV-1 RNA, <=100000,n=294, 282: number analyzed (Participants) | 294 | 282
  Baseline plasma HIV-1 RNA, <=100000,n=294, 282 | 88 | 91
  Baseline plasma HIV-1 RNA, >100000,n=66, 77: number analyzed (Participants) | 66 | 77
  Baseline plasma HIV-1 RNA, >100000,n=66, 77 | 86 | 84
  Race, White, n=240,252: number analyzed (Participants) | 240 | 252
  Race, White, n=240,252 | 92 | 91
  Race, African American/African H., n=51, 35: number analyzed (Participants) | 51 | 35
  Race, African American/African H., n=51, 35 | 69 | 86
  Race, Asian, n=34, 30: number analyzed (Participants) | 34 | 30
  Race, Asian, n=34, 30 | 88 | 90
  Race, Other, n=35, 42: number analyzed (Participants) | 35 | 42
  Race, Other, n=35, 42 | 89 | 83

54. Secondary Outcome: Percentage of Participants by Subgroups (by Age, Gender, Baseline CD4+ Cell Count Baseline HIV-1 RNA, Race) With Plasma HIV-1 RNA <50 c/mL at Week 144
Description: as for outcome 53
Time Frame: Week 144
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 360 | 359
Percentage of participants
  Baseline CD4+ cell count, <=200,n=32, 26: number analyzed (Participants) | 32 | 26
  Baseline CD4+ cell count, <=200,n=32, 26 | 75 | 69
  Baseline CD4+ cell count, >200,n=328,333: number analyzed (Participants) | 328 | 333
  Baseline CD4+ cell count, >200,n=328,333 | 85 | 86
  Female, n=54, 46: number analyzed (Participants) | 54 | 46
  Female, n=54, 46 | 78 | 83
  Male, n=306, 313: number analyzed (Participants) | 306 | 313
  Male, n=306, 313 | 85 | 85
  Age, <35,n= 209, 203: number analyzed (Participants) | 209 | 203
  Age, <35,n= 209, 203 | 83 | 83
  Age, 35 to <50,n=115, 122: number analyzed (Participants) | 115 | 122
  Age, 35 to <50,n=115, 122 | 86 | 85
  Age, >=50, n=36, 34: number analyzed (Participants) | 36 | 34
  Age, >=50, n=36, 34 | 83 | 88
  Baseline plasma HIV-1 RNA, <=100000,n=294, 282: number analyzed (Participants) | 294 | 282
  Baseline plasma HIV-1 RNA, <=100000,n=294, 282 | 84 | 85
  Baseline plasma HIV-1 RNA, >100000,n=66, 77: number analyzed (Participants) | 66 | 77
  Baseline plasma HIV-1 RNA, >100000,n=66, 77 | 86 | 81
  Race, White, n=240,252: number analyzed (Participants) | 240 | 252
  Race, White, n=240,252 | 88 | 87
  Race, African American/African H., n=51, 35: number analyzed (Participants) | 51 | 35
  Race, African American/African H., n=51, 35 | 65 | 74
  Race, Asian, n=34, 30: number analyzed (Participants) | 34 | 30
  Race, Asian, n=34, 30 | 85 | 83
  Race, Other, n=35, 42: number analyzed (Participants) | 35 | 42
  Race, Other, n=35, 42 | 89 | 79

55. Secondary Outcome: Changes From Baseline in CD4+ Cell Counts at Week 24 by Subgroups
Description: CD4+ cells are type of white blood cells that fight infection and as HIV infection progresses, the number of these cells declines. Blood samples were collected at specified time points to assess CD4+. It was evaluated by flow cytometry. Baseline value is the latest pre-dose assessment (Day 1). Change from Baseline was defined as value at the indicated time point minus Baseline value. Adjusted mean and standard error is presented for subgroups (Baseline plasma HIV-1 RNA, Baseline CD4+ cell count, Age group, Gender and race). For each subgroup, adjusted mean is the estimated mean change from Baseline in each arm calculated from ANCOVA model adjusting for the following covariates/factors: treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, subgroup, and treatment and relevant subgroup interaction. For CD4+ cell count subgroup, Baseline CD4+ cell count group is included as a factor only.
Time Frame: Baseline (Day 1) and Week 24
Population: as for outcome 6
Measure: Mean (Standard Error); unit: Cells/mm^3
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 360 | 359
Cells/mm^3
  Baseline plasma HIV-1 RNA,<=100000, n=283,273: number analyzed (Participants) | 283 | 273
  Baseline plasma HIV-1 RNA,<=100000, n=283,273 | 186.01 (9.948) | 148.21 (10.134)
  Baseline plasma HIV-1 RNA,>100000, n=66,72: number analyzed (Participants) | 66 | 72
  Baseline plasma HIV-1 RNA,>100000, n=66,72 | 193.90 (20.811) | 220.71 (19.814)
  Baseline CD4+ cell count,<=200, n=29, 26: number analyzed (Participants) | 29 | 26
  Baseline CD4+ cell count,<=200, n=29, 26 | 167.95 (31.308) | 106.23 (32.990)
  Baseline CD4+ cell count,>200, n=320, 319: number analyzed (Participants) | 320 | 319
  Baseline CD4+ cell count,>200, n=320, 319 | 189.91 (9.362) | 167.35 (9.362)
  Age group, <35,n= 201, 193: number analyzed (Participants) | 201 | 193
  Age group, <35,n= 201, 193 | 190.12 (11.829) | 151.13 (12.050)
  Age group-1, 35 to <50, n=113, 119: number analyzed (Participants) | 113 | 119
  Age group-1, 35 to <50, n=113, 119 | 180.50 (15.733) | 190.40 (15.404)
  Age group-1, >=50, n=35, 33: number analyzed (Participants) | 35 | 33
  Age group-1, >=50, n=35, 33 | 198.74 (28.411) | 133.21 (29.120)
  Female, n=52, 42: number analyzed (Participants) | 52 | 42
  Female, n=52, 42 | 213.58 (23.225) | 153.92 (25.910)
  Male, n=297, 303: number analyzed (Participants) | 297 | 303
  Male, n=297, 303 | 183.41 (9.719) | 164.18 (9.631)
  Race group, White, n=236, 243: number analyzed (Participants) | 236 | 243
  Race group, White, n=236, 243 | 186.48 (10.932) | 167.44 (10.790)
  Race group, African Am/African H., n=48, 34: number analyzed (Participants) | 48 | 34
  Race group, African Am/African H., n=48, 34 | 195.18 (24.222) | 151.93 (28.784)
  Race group, Asian, n=33, 28: number analyzed (Participants) | 33 | 28
  Race group, Asian, n=33, 28 | 154.03 (29.438) | 141.24 (31.703)
  Race group, Other, n=32, 40: number analyzed (Participants) | 32 | 40
  Race group, Other, n=32, 40 | 222.21 (29.681) | 160.20 (26.627)
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = 37.80, 95% CI 2-sided [9.98 to 65.62] — Baseline plasma HIV-1 RNA,<=100000. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, Baseline plasma HIV-1 RNA, and treatment and relevant Baseline plasma HIV-1 RNA interaction
Statistical Analysis 2: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = -26.81, 95% CI 2-sided [-82.72 to 29.10] — Baseline plasma HIV-1 RNA,>100000. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, Baseline plasma HIV-1 RNA, and treatment and Baseline plasma HIV-1 RNA interaction
Statistical Analysis 3: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = 61.72, 95% CI 2-sided [-26.94 to 150.39] — Baseline CD4+ cell count,<=200. Following covariates were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, and treatment and Baseline CD4+ cell count interaction
Statistical Analysis 4: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = 22.57, 95% CI 2-sided [-3.42 to 48.55] — Baseline CD4+ cell count,>200. Following covariates were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, and treatment and Baseline CD4+ cell count interaction
Statistical Analysis 5: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = 38.99, 95% CI 2-sided [5.88 to 72.09] — Age Group,<35. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, age, and treatment and age interaction
Statistical Analysis 6: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = -9.90, 95% CI 2-sided [-53.10 to 33.30] — Age Group,35 to <50. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, age, and treatment and age interaction
Statistical Analysis 7: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = 65.53, 95% CI 2-sided [-14.43 to 145.50] — Age Group,>=50. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, age, and treatment and age interaction
Statistical Analysis 8: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = 59.66, 95% CI 2-sided [-8.62 to 127.94] — Female. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, gender, and treatment and gender interaction
Statistical Analysis 9: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = 19.23, 95% CI 2-sided [-7.65 to 46.10] — Male. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, gender, and treatment and gender interaction
Statistical Analysis 10: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = 19.04, 95% CI 2-sided [-11.06 to 49.13] — Race group-white. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, race, and treatment and race interaction
Statistical Analysis 11: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = 43.25, 95% CI 2-sided [-30.59 to 117.09] — Race group-African Am/African H. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, race, and treatment and race interaction
Statistical Analysis 12: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = 12.80, 95% CI 2-sided [-72.14 to 97.73] — Race group-Asian. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, race, and treatment and race interaction
Statistical Analysis 13: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = 62.01, 95% CI 2-sided [-16.09 to 140.12] — Race group-Other. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, race, and treatment and race interaction

56. Secondary Outcome: Changes From Baseline in CD4+ Cell Counts at Week 48 by Subgroups
Description: CD4+ cells are type of white blood cells that fight infection and as HIV infection progresses, the number of these cells declines. Blood samples were collected at specified time points to assess CD4+. It was evaluated by flow cytometry. Baseline value is the latest pre-dose assessment (Day 1). Change from Baseline was defined as value at the indicated time point minus Baseline value. Adjusted mean and standard error is presented for subgroups (Baseline plasma HIV-1 RNA, Baseline CD4+ cell count, Age group, Gender and race). For each subgroup, adjusted mean is the estimated mean change from Baseline in each arm calculated from Analysis of Covariance (ANCOVA) model adjusting for the following covariates/factors: treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, subgroup, and treatment and relevant subgroup interaction. For CD4+ cell count subgroup, Baseline CD4+ cell count group is included as a factor only.
Time Frame: Baseline (Day 1) and Week 48
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Cells/mm^3
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 360 | 359
Cells/mm^3
  Baseline plasma HIV-1 RNA,<=100000, n=273,271: number analyzed (Participants) | 273 | 271
  Baseline plasma HIV-1 RNA,<=100000, n=273,271 | 215.6 (10.67) | 208.7 (10.71)
  Baseline plasma HIV-1 RNA,>100000, n=64,69: number analyzed (Participants) | 64 | 69
  Baseline plasma HIV-1 RNA,>100000, n=64,69 | 261.8 (22.27) | 248.7 (21.30)
  Baseline CD4+ cell count,<=200, n=28, 25: number analyzed (Participants) | 28 | 25
  Baseline CD4+ cell count,<=200, n=28, 25 | 210.9 (33.42) | 153.2 (35.29)
  Baseline CD4+ cell count,>200, n=309, 315: number analyzed (Participants) | 309 | 315
  Baseline CD4+ cell count,>200, n=309, 315 | 225.8 (10.00) | 221.7 (9.89)
  Age group-1, <35,n= 193, 191: number analyzed (Participants) | 193 | 191
  Age group-1, <35,n= 193, 191 | 234.2 (12.67) | 201.7 (12.72)
  Age group-1, 35 to <50, n=112, 117: number analyzed (Participants) | 112 | 117
  Age group-1, 35 to <50, n=112, 117 | 212.7 (16.59) | 244.2 (16.31)
  Age group-1, >=50, n=32, 32: number analyzed (Participants) | 32 | 32
  Age group-1, >=50, n=32, 32 | 209.1 (31.20) | 203.9 (31.06)
  Age group-2, <50,n= 305, 308: number analyzed (Participants) | 305 | 308
  Age group-2, <50,n= 305, 308 | 226.4 (10.09) | 217.8 (10.03)
  Age group-2, >=50, n= 32, 32: number analyzed (Participants) | 32 | 32
  Age group-2, >=50, n= 32, 32 | 208.5 (31.27) | 204.1 (31.14)
  Female, n=48, 41: number analyzed (Participants) | 48 | 41
  Female, n=48, 41 | 236.2 (25.35) | 263.6 (27.50)
  Male, n=289, 299: number analyzed (Participants) | 289 | 299
  Male, n=289, 299 | 222.8 (10.33) | 210.0 (10.17)
  Race group, White, n=230, 244: number analyzed (Participants) | 230 | 244
  Race group, White, n=230, 244 | 225.5 (11.62) | 214.2 (11.30)
  Race group, African Am/African H., n=42, 31: number analyzed (Participants) | 42 | 31
  Race group, African Am/African H., n=42, 31 | 201.2 (27.16) | 239.0 (31.64)
  Race group, Asian, n=33, 27: number analyzed (Participants) | 33 | 27
  Race group, Asian, n=33, 27 | 204.9 (30.90) | 189.3 (33.88)
  Race group, Other, n=32, 38: number analyzed (Participants) | 32 | 38
  Race group, Other, n=32, 38 | 270.2 (31.15) | 232.6 (28.67)
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = 6.9, 95% CI 2-sided [-22.7 to 36.6] — [estimate comment as in outcome 55, analysis 1]
Statistical Analysis 2: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = 13.2, 95% CI 2-sided [-46.8 to 73.2] — [estimate comment as in outcome 55, analysis 2]
Statistical Analysis 3: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = 57.7, 95% CI 2-sided [-37.2 to 152.5] — [estimate comment as in outcome 55, analysis 3]
Statistical Analysis 4: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = 4.1, 95% CI 2-sided [-23.5 to 31.7] — [estimate comment as in outcome 55, analysis 4]
Statistical Analysis 5: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = 32.5, 95% CI 2-sided [-2.7 to 67.7] — Age Group-1,<35. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, age, and treatment and age interaction
Statistical Analysis 6: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = -31.5, 95% CI 2-sided [-77.1 to 14.2] — Age Group-1,35 to <50. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, age, and treatment and age interaction
Statistical Analysis 7: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = 5.2, 95% CI 2-sided [-81.4 to 91.8] — Age Group-1,>=50. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, age, and treatment and age interaction
Statistical Analysis 8: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = 8.6, 95% CI 2-sided [-19.4 to 36.5] — Age Group-2, <50. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, age, and treatment and age interaction
Statistical Analysis 9: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = 4.5, 95% CI 2-sided [-82.3 to 91.3] — Age Group-2, >=50. Following covariates/factors were adjusted: Treatment, Baseline plasma HIV-1 RNA (factor), Baseline CD4+ cell count, age, and treatment and age interaction
Statistical Analysis 10: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = -27.3, 95% CI 2-sided [-100.8 to 46.1] — [estimate comment as in outcome 55, analysis 8]
Statistical Analysis 11: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = 12.8, 95% CI 2-sided [-15.7 to 41.2] — [estimate comment as in outcome 55, analysis 9]
Statistical Analysis 12: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = 11.3, 95% CI 2-sided [-20.4 to 43.1] — [estimate comment as in outcome 55, analysis 10]
Statistical Analysis 13: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = -37.8, 95% CI 2-sided [-119.6 to 44.0] — [estimate comment as in outcome 55, analysis 11]
Statistical Analysis 14: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = 15.6, 95% CI 2-sided [-74.4 to 105.7] — [estimate comment as in outcome 55, analysis 12]
Statistical Analysis 15: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = 37.6, 95% CI 2-sided [-45.4 to 120.5] — [estimate comment as in outcome 55, analysis 13]

57. Secondary Outcome: Changes From Baseline in CD4+ Cell Counts at Week 96 by Subgroups
Description: as for outcome 55
Time Frame: Baseline (Day 1) and Week 96
Population: as for outcome 6
Measure: Mean (Standard Error); unit: Cells/mm^3
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 360 | 359
Cells/mm^3
  Baseline plasma HIV-1 RNA,<=100000, n=259,260: number analyzed (Participants) | 259 | 260
  Baseline plasma HIV-1 RNA,<=100000, n=259,260 | 257.9 (12.47) | 257.5 (12.45)
  Baseline plasma HIV-1 RNA,>100000, n=59,67: number analyzed (Participants) | 59 | 67
  Baseline plasma HIV-1 RNA,>100000, n=59,67 | 312.1 (26.37) | 297.4 (24.59)
  Baseline CD4+ cell count,<=200, n=25, 23: number analyzed (Participants) | 25 | 23
  Baseline CD4+ cell count,<=200, n=25, 23 | 229.4 (40.41) | 202.9 (42.00)
  Baseline CD4+ cell count,>200, n=293, 304: number analyzed (Participants) | 293 | 304
  Baseline CD4+ cell count,>200, n=293, 304 | 272.3 (11.73) | 269.4 (11.50)
  Age group-1, <35,n= 186, 187: number analyzed (Participants) | 186 | 187
  Age group-1, <35,n= 186, 187 | 266.0 (14.74) | 257.7 (14.68)
  Age group-1, 35 to <50, n=101, 110: number analyzed (Participants) | 101 | 110
  Age group-1, 35 to <50, n=101, 110 | 273.6 (19.95) | 286.8 (19.22)
  Age group-1, >=50, n=31, 30: number analyzed (Participants) | 31 | 30
  Age group-1, >=50, n=31, 30 | 265.8 (36.14) | 233.1 (36.61)
  Female, n=44, 40: number analyzed (Participants) | 44 | 40
  Female, n=44, 40 | 312.7 (30.12) | 307.6 (31.67)
  Male, n=274, 287: number analyzed (Participants) | 274 | 287
  Male, n=274, 287 | 261.4 (12.07) | 259.3 (11.81)
  Race group, White, n=221, 234: number analyzed (Participants) | 221 | 234
  Race group, White, n=221, 234 | 272.1 (13.49) | 258.3 (13.14)
  Race group, African Am/African H., n=35, 30: number analyzed (Participants) | 35 | 30
  Race group, African Am/African H., n=35, 30 | 246.3 (33.90) | 303.7 (36.61)
  Race group, Asian, n=31, 27: number analyzed (Participants) | 31 | 27
  Race group, Asian, n=31, 27 | 224.0 (36.31) | 264.0 (38.57)
  Race group, Other, n=31, 36: number analyzed (Participants) | 31 | 36
  Race group, Other, n=31, 36 | 312.0 (36.01) | 278.9 (33.56)
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = 0.5, 95% CI 2-sided [-34.1 to 35.0] — [estimate comment as in outcome 55, analysis 1]
Statistical Analysis 2: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = 14.7, 95% CI 2-sided [-55.6 to 84.9] — [estimate comment as in outcome 55, analysis 2]
Statistical Analysis 3: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = 26.5, 95% CI 2-sided [-87.3 to 140.3] — [estimate comment as in outcome 55, analysis 3]
Statistical Analysis 4: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = 2.8, 95% CI 2-sided [-29.4 to 35.1] — [estimate comment as in outcome 55, analysis 4]
Statistical Analysis 5: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = 8.3, 95% CI 2-sided [-32.5 to 49.1] — [estimate comment as in outcome 55, analysis 5]
Statistical Analysis 6: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = -13.3, 95% CI 2-sided [-67.6 to 41.1] — [estimate comment as in outcome 55, analysis 6]
Statistical Analysis 7: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = 32.7, 95% CI 2-sided [-68.5 to 133.9] — [estimate comment as in outcome 55, analysis 7]
Statistical Analysis 8: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = 5.1, 95% CI 2-sided [-80.7 to 90.8] — [estimate comment as in outcome 55, analysis 8]
Statistical Analysis 9: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = 2.1, 95% CI 2-sided [-31.1 to 35.3] — [estimate comment as in outcome 55, analysis 9]
Statistical Analysis 10: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = 13.7, 95% CI 2-sided [-23.2 to 50.6] — [estimate comment as in outcome 55, analysis 10]
Statistical Analysis 11: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = -57.4, 95% CI 2-sided [-155.3 to 40.4] — [estimate comment as in outcome 55, analysis 11]
Statistical Analysis 12: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = -40.1, 95% CI 2-sided [-144.2 to 64.0] — [estimate comment as in outcome 55, analysis 12]
Statistical Analysis 13: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; Mean Difference (Net) = 33.1, 95% CI 2-sided [-63.3 to 129.6] — [estimate comment as in outcome 55, analysis 13]

58. Secondary Outcome: Changes From Baseline in CD4+ Cell Counts at Week 144 by Subgroups
Description: as for outcome 55
Time Frame: Baseline (Day 1) and Week 144
Population: as for outcome 6
Measure: Mean (Standard Error); unit: Cells/mm^3
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 360 | 359
Cells/mm^3
  Baseline plasma HIV-1 RNA,<=100000, n=241,234: number analyzed (Participants) | 241 | 234
  Baseline plasma HIV-1 RNA,<=100000, n=241,234 | 286.8 (14.36) | 277.8 (14.58)
  Baseline plasma HIV-1 RNA,>100000, n=55,58: number analyzed (Participants) | 55 | 58
  Baseline plasma HIV-1 RNA,>100000, n=55,58 | 338.2 (30.34) | 354.7 (29.35)
  Baseline CD4+ cell count,<=200, n=25, 19: number analyzed (Participants) | 25 | 19
  Baseline CD4+ cell count,<=200, n=25, 19 | 264.8 (44.91) | 208.9 (51.25)
  Baseline CD4+ cell count,>200, n=271, 273: number analyzed (Participants) | 271 | 273
  Baseline CD4+ cell count,>200, n=271, 273 | 300.3 (13.54) | 297.9 (13.48)
  Age group, <35,n=171, 159: number analyzed (Participants) | 171 | 159
  Age group, <35,n=171, 159 | 302.9 (17.05) | 277.1 (17.65)
  Age group-1, 35 to <50, n=95, 103: number analyzed (Participants) | 95 | 103
  Age group-1, 35 to <50, n=95, 103 | 292.8 (22.82) | 329.2 (22.02)
  Age group-1, >=50, n=30, 30: number analyzed (Participants) | 30 | 30
  Age group-1, >=50, n=30, 30 | 274.1 (40.71) | 250.0 (40.60)
  Female, n=40, 37: number analyzed (Participants) | 40 | 37
  Female, n=40, 37 | 355.0 (34.93) | 381.8 (36.37)
  Male, n=256, 255: number analyzed (Participants) | 256 | 255
  Male, n=256, 255 | 287.7 (13.81) | 279.6 (13.85)
  Race group, White, n=202, 211: number analyzed (Participants) | 202 | 211
  Race group, White, n=202, 211 | 300.0 (15.61) | 296.5 (15.29)
  Race group, African Am/African H., n=34, 24: number analyzed (Participants) | 34 | 24
  Race group, African Am/African H., n=34, 24 | 256.4 (38.04) | 377.6 (45.25)
  Race group, Asian, n=29, 25: number analyzed (Participants) | 29 | 25
  Race group, Asian, n=29, 25 | 258.5 (41.57) | 245.4 (44.36)
  Race group, Other, n=31, 32: number analyzed (Participants) | 31 | 32
  Race group, Other, n=31, 32 | 355.0 (39.84) | 240.7 (39.35)
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; Mean Difference (Net) = 9.1, 95% CI 2-sided [-31.1 to 49.2] — [estimate comment as in outcome 55, analysis 1]
Statistical Analysis 2: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; Mean Difference (Net) = -16.6, 95% CI 2-sided [-98.9 to 65.8] — [estimate comment as in outcome 55, analysis 2]
Statistical Analysis 3: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; Mean Difference (Net) = 56.0, 95% CI 2-sided [-77.2 to 189.1] — [estimate comment as in outcome 55, analysis 3]
Statistical Analysis 4: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; Mean Difference (Net) = 2.4, 95% CI 2-sided [-35.2 to 39.9] — [estimate comment as in outcome 55, analysis 4]
Statistical Analysis 5: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; Mean Difference (Net) = 25.8, 95% CI 2-sided [-22.3 to 74.0] — [estimate comment as in outcome 55, analysis 5]
Statistical Analysis 6: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; Mean Difference (Net) = -36.4, 95% CI 2-sided [-98.6 to 25.8] — [estimate comment as in outcome 55, analysis 6]
Statistical Analysis 7: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; Mean Difference (Net) = 24.1, 95% CI 2-sided [-89.0 to 137.2] — [estimate comment as in outcome 55, analysis 7]
Statistical Analysis 8: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; Mean Difference (Net) = -26.9, 95% CI 2-sided [-125.9 to 72.2] — [estimate comment as in outcome 55, analysis 8]
Statistical Analysis 9: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; Mean Difference (Net) = 8.1, 95% CI 2-sided [-30.3 to 46.5] — [estimate comment as in outcome 55, analysis 9]
Statistical Analysis 10: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; Mean Difference (Net) = 3.5, 95% CI 2-sided [-39.4 to 46.3] — [estimate comment as in outcome 55, analysis 10]
Statistical Analysis 11: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; Mean Difference (Net) = -121.2, 95% CI 2-sided [-237.2 to -5.1] — [estimate comment as in outcome 55, analysis 11]
Statistical Analysis 12: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; Mean Difference (Net) = 13.1, 95% CI 2-sided [-106.4 to 132.6] — [estimate comment as in outcome 55, analysis 12]
Statistical Analysis 13: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; Mean Difference (Net) = 114.3, 95% CI 2-sided [4.6 to 224.0] — [estimate comment as in outcome 55, analysis 13]

59. Secondary Outcome: Change From Baseline in European Quality of Life [EuroQoL] - 5 Dimensions - 5 Levels (EQ-5D-5L) Utility Score at Weeks 4, 24, 48
Description: EQ-5D-5L questionnaire provides a profile of participant function and a global health state rating. The five-item measure has 1 question assessing each of 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression and 5 levels for each dimension including 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems and 5=extreme problems. The health state is defined by combining the levels of answers from each of the 5 questions. Each health state is referred to in terms of a 5 digit code. Health state 5 digit code is translated into utility score, which is valued up to 1 (perfect health) with lower values meaning worse state. EQ-5D-5L utility score ranges from -0.281 to 1. Higher scores indicate better health. MMRM was run on LOCF dataset. Baseline was the latest pre-dose assessment and change from Baseline=post-dose value minus Baseline value.
Time Frame: Baseline (Day 1) and Weeks 4, 24, 48
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 360 | 359
Scores on a scale
  Week 4, n=359, 355: number analyzed (Participants) | 359 | 355
  Week 4, n=359, 355 | 0.0111 (0.00326) | 0.0130 (0.00510)
  Week 24, n=360, 358: number analyzed (Participants) | 360 | 358
  Week 24, n=360, 358 | 0.0207 (0.00310) | 0.0203 (0.00347)
  Week 48, n=360, 358: number analyzed (Participants) | 360 | 358
  Week 48, n=360, 358 | 0.0189 (0.00362) | 0.0208 (0.00342)
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p = 0.759, MMRM; Mean Difference (Net) = -0.0019, 95% CI 2-sided [-0.0137 to 0.0100] — Week 4. Covariates adjusted: Treatment, Baseline plasma HIV-1 RNA , Baseline CD4+ cell count , and Baseline EQ-5D utility, treatment*visit and Baseline EQ-5D utility*visit as factors and covariate, with visit as the repeated factor
Statistical Analysis 2: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p = 0.943, MMRM; Mean Difference (Net) = 0.0003, 95% CI 2-sided [-0.0088 to 0.0095] — Week 24. Covariates adjusted: Treatment, Baseline plasma HIV-1 RNA , Baseline CD4+ cell count , and Baseline EQ-5D utility, treatment*visit and Baseline EQ-5D utility*visit as factors and covariate, with visit as the repeated factor
Statistical Analysis 3: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p = 0.703, MMRM; Mean Difference (Net) = -0.0019, 95% CI 2-sided [-0.0117 to 0.0079] — Week 48. Covariates adjusted: Treatment, Baseline plasma HIV-1 RNA , Baseline CD4+ cell count , and Baseline EQ-5D utility, treatment*visit and Baseline EQ-5D utility*visit as factors and covariate, with visit as the repeated factor

60. Secondary Outcome: Change From Baseline in EQ-5D-5L Utility Score at Week 96
Description: EQ-5D-5L questionnaire provides a profile of participant function and a global health state rating. The five-item measure has 1 question assessing each of 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression and 5 levels for each dimension including 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems and 5=extreme problems. The health state is defined by combining the levels of answers from each of the 5 questions. Each health state is referred to in terms of a 5 digit code. Health state 5 digit code is translated into utility score, which is valued up to 1 (perfect health) with lower values meaning worse state. EQ-5D-5L utility score ranges from -0.281 to 1. Higher scores indicate better health. MMRM was run on LOCF dataset. Baseline was the latest pre-dose assessment and change from Baseline=post-dose value minus Baseline value. Adjusted mean and standard error is presented.
Time Frame: Baseline (Day 1) and Week 96
Population: ITT-E Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 360 | 358
Scores on a scale | 0.0168 (0.00339) | 0.0171 (0.00424)
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p = 0.957, MMRM; Mean Difference (Net) = -0.0003, 95% CI 2-sided [-0.0110 to 0.0104] — Week 96. Covariates adjusted: Treatment, Baseline plasma HIV-1 RNA, Baseline CD4+ cell count, and Baseline EQ-5D utility, treatment*visit and Baseline EQ-5D utility*visit as factors and covariate, with visit as the repeated factor

61. Secondary Outcome: Change From Baseline in EQ-5D-5L Utility Score at Week 144
Description: as for outcome 60
Time Frame: Baseline (Day 1) and Week 144
Population: ITT-E Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 360 | 358
Scores on a scale | 0.0210 (0.00346) | 0.0131 (0.00441)
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; p = 0.162, MMRM; Mean Difference (Net) = 0.0079, 95% CI 2-sided [-0.0032 to 0.0189] — Week 144. Covariates adjusted: Treatment, Baseline plasma HIV-1 RNA, Baseline CD4+ cell count, and Baseline EQ-5D utility, treatment*visit and Baseline EQ-5D utility*visit as factors and covariate, with visit as the repeated factor

62. Secondary Outcome: Change From Baseline in EuroQol - 5 Dimensions - 5 Levels (EQ-5D-5L) Thermometer Scores at Weeks 4, 24, 48
Description: EQ-5D-5L questionnaire provided a profile of participant function and a global health state rating. The five-item measure has one question assessing each of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression and 5 levels for each dimension including 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems and 5=extreme problems. EQ-5D-5L included EQ visual Analogue scale (EQ VAS) 'Thermometer' which provided Self-rated current health status. Score ranges from 0 (worst imaginable health state) to 100 (best imaginable health state). MMRM was run on the LOCF dataset, using the observed margins (OM) option. Baseline was the latest pre-dose assessment value and change from Baseline=post-dose value minus Baseline value.
Time Frame: Baseline (Day 1) and Weeks 4, 24, 48
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 360 | 359
Scores on a scale
  Week 4, n=358, 355: number analyzed (Participants) | 358 | 355
  Week 4, n=358, 355 | 1.8 (0.50) | 3.1 (0.41)
  Week 24, n=359, 358: number analyzed (Participants) | 359 | 358
  Week 24, n=359, 358 | 3.9 (0.43) | 4.5 (0.48)
  Week 48, n=359, 358: number analyzed (Participants) | 359 | 358
  Week 48, n=359, 358 | 4.0 (0.43) | 4.6 (0.48)
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p = 0.045, MMRM; Mean Difference (Net) = -1.3, 95% CI 2-sided [-2.6 to 0.0] — Week 4. Covariates adjusted: Treatment, Baseline plasma HIV-1 RNA, Baseline CD4+ cell count and Baseline EQ-5D utility, treatment*visit and Baseline EQ-5D utility*visit as factors and covariate, with visit as the repeated factor
Statistical Analysis 2: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p = 0.358, MMRM; Mean Difference (Net) = -0.6, 95% CI 2-sided [-1.9 to 0.7] — Week 24. Covariates adjusted: Treatment, Baseline plasma HIV-1 RNA, Baseline CD4+ cell count and Baseline EQ-5D utility, treatment*visit and Baseline EQ-5D utility*visit as factors and covariate, with visit as the repeated factor
Statistical Analysis 3: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p = 0.328, MMRM; Mean Difference (Net) = -0.6, 95% CI 2-sided [-1.9 to 0.6] — Week 48. Covariates adjusted: Treatment, Baseline plasma HIV-1 RNA, Baseline CD4+ cell count, and Baseline EQ-5D utility, treatment*visit and Baseline EQ-5D utility*visit as factors and covariate, with visit as the repeated factor

63. Secondary Outcome: Change From Baseline in EQ-5D-5L Thermometer Scores at Week 96
Description: EQ-5D-5L questionnaire provided a profile of participant function and a global health state rating. The five-item measure has one question assessing each of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression and 5 levels for each dimension including 1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems and 5=extreme problems. EQ-5D-5L included EQ visual Analogue scale (EQ VAS) 'Thermometer' which provided Self-rated current health status. Score ranges from 0 (worst imaginable health state) to 100 (best imaginable health state). MMRM was run on the LOCF dataset, using the observed margins (OM) option. Baseline was the latest pre-dose assessment value and change from Baseline=post-dose value minus Baseline value. Adjusted mean and standard error is presented.
Time Frame: Baseline (Day 1) and Week 96
Population: ITT-E Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | DTG + 3TC - Double-blind Phase | DTG + TDF/FTC - Double-blind Phase
Number analyzed (Participants) | 359 | 358
Scores on a scale | 4.4 (0.45) | 5.1 (0.52)
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase vs DTG + TDF/FTC - Double-blind Phase; Test type: Other; p = 0.318, MMRM; Mean Difference (Net) = -0.7, 95% CI 2-sided [-2.1 to 0.7] — Week 96. Covariates adjusted: Treatment, Baseline plasma HIV-1 RNA, Baseline CD4+ cell count and Baseline EQ-5D utility, treatment*visit and Baseline EQ-5D utility*visit as factors and covariate, with visit as the repeated factor

64. Secondary Outcome: Change From Baseline in EQ-5D-5L Thermometer Scores at Week 144
Description: as for outcome 63
Time Frame: Baseline (Day 1) and Week 144
Population: ITT-E Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase
Number analyzed (Participants) | 359 | 358
Scores on a scale | 4.8 (0.44) | 4.5 (0.51)
Statistical Analysis 1: Comparison: DTG + 3TC - Double-blind Phase + Open-label Phase vs DTG + TDF/FTC - Double-blind Phase + Open-label Phase; Test type: Other; p = 0.674, MMRM; Mean Difference (Net) = 0.3, 95% CI 2-sided [-1.0 to 1.6] — Week 144. Covariates adjusted: Treatment, Baseline plasma HIV-1 RNA, Baseline CD4+ cell count and Baseline EQ-5D utility, treatment*visit and Baseline EQ-5D utility*visit as factors and covariate, with visit as the repeated factor

ADVERSE EVENTS:
Time Frame: All-cause mortality, SAEs and non-SAEs were collected up to Week 148 in Double-blind Phase + Open-label Phase and from Week 148 to Week 280 in Continuation Phase
Description: All-cause mortality, SAEs and non-SAEs were reported for the Safety Population for the Double-blind Phase and Double-blind Phase + Open-label Phase. Safety-Continuation Population was used for the Continuation Phase (which comprised of all participants who received at least 1 dose of study treatment after entering the Continuation Phase).
Arm/Group | DTG + 3TC - Double-blind Phase + Open-label Phase | DTG + TDF/FTC - Double-blind Phase + Open-label Phase | DTG + 3TC - Continuation Phase
All-Cause Mortality (participants affected / at risk) | 2/360 | 1/359 | 0/252
Serious Adverse Events (participants affected / at risk) | 39/360 | 47/359 | 9/252
Other Adverse Events (participants affected / at risk) | 273/360 | 276/359 | 45/252
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTG + 3TC - Double-blind Phase + Open-label Phase (N=360) | DTG + TDF/FTC - Double-blind Phase + Open-label Phase (N=359) | DTG + 3TC - Continuation Phase (N=252)
Hepatitis A (Infections and infestations) | 3 (3) | 3 (3) | 1 (1)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3) | 0 (0)
Suicide attempt (Psychiatric disorders) | 5 (5) | 2 (3) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 4 (6) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Acute hepatitis C (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 3 (3) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Alcoholic psychosis (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Anal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bacterial colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fracture of penis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Ophthalmic vein thrombosis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Penetrating abdominal trauma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 2 (4) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tuberculous pleurisy (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Urethral meatus stenosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Chronic tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hepatitis C (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Jarisch-Herxheimer reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Substance-induced psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis orbital (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis cryptosporidial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Labyrinthitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Shigella infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Syphilis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Traumatic arthritis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Migraine with aura (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gallbladder rupture (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DTG + 3TC - Double-blind Phase + Open-label Phase (N=360) | DTG + TDF/FTC - Double-blind Phase + Open-label Phase (N=359) | DTG + 3TC - Continuation Phase (N=252)
Diarrhoea (Gastrointestinal disorders) | 49 (55) | 53 (61) | 0 (0)
Nasopharyngitis (Infections and infestations) | 44 (59) | 69 (103) | 0 (0)
Headache (Nervous system disorders) | 33 (49) | 44 (60) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 47 (75) | 28 (44) | 7 (7)
Nausea (Gastrointestinal disorders) | 16 (17) | 31 (33) | 0 (0)
Pharyngitis (Infections and infestations) | 24 (31) | 33 (35) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 27 (32) | 23 (30) | 0 (0)
Insomnia (Psychiatric disorders) | 17 (17) | 23 (28) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 (21) | 25 (26) | 0 (0)
Influenza (Infections and infestations) | 16 (17) | 25 (27) | 0 (0)
Syphilis (Infections and infestations) | 26 (30) | 30 (34) | 10 (11)
Anxiety (Psychiatric disorders) | 17 (17) | 18 (19) | 0 (0)
Dizziness (Nervous system disorders) | 9 (11) | 18 (20) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 17 (21) | 16 (17) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 14 (20) | 12 (19) | 8 (10)
Abdominal pain (Gastrointestinal disorders) | 9 (10) | 17 (17) | 0 (0)
Bronchitis (Infections and infestations) | 12 (14) | 21 (24) | 0 (0)
Gastroenteritis (Infections and infestations) | 21 (21) | 20 (25) | 6 (6)
Haemorrhoids (Gastrointestinal disorders) | 16 (17) | 12 (12) | 0 (0)
Tonsillitis (Infections and infestations) | 13 (14) | 9 (13) | 0 (0)
Constipation (Gastrointestinal disorders) | 9 (9) | 14 (14) | 0 (0)
Fatigue (General disorders) | 10 (13) | 9 (9) | 0 (0)
Gonorrhoea (Infections and infestations) | 12 (14) | 12 (15) | 0 (0)
Influenza like illness (General disorders) | 16 (20) | 11 (14) | 0 (0)
Toothache (Gastrointestinal disorders) | 7 (8) | 14 (15) | 0 (0)
Vomiting (Gastrointestinal disorders) | 11 (11) | 11 (12) | 0 (0)
Chlamydial infection (Infections and infestations) | 10 (13) | 13 (13) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 15 (15) | 0 (0)
Depression (Psychiatric disorders) | 12 (14) | 13 (16) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 10 (13) | 13 (16) | 0 (0)
Pyrexia (General disorders) | 11 (11) | 9 (12) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 28 (29) | 20 (20) | 0 (0)
Rhinitis (Infections and infestations) | 5 (6) | 16 (18) | 0 (0)
Dysuria (Renal and urinary disorders) | 10 (10) | 3 (3) | 0 (0)
Genital herpes (Infections and infestations) | 4 (4) | 10 (14) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 15 (15)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 7 (8)
Anal chlamydia infection (Infections and infestations) | 10 (12) | 16 (21) | 0 (0)
Sinusitis (Infections and infestations) | 12 (14) | 12 (13) | 0 (0)
Urinary tract infection (Infections and infestations) | 11 (14) | 9 (12) | 0 (0)
Proctitis gonococcal (Infections and infestations) | 9 (12) | 9 (11) | 0 (0)
Respiratory tract infection (Infections and infestations) | 10 (12) | 8 (10) | 0 (0)
Secondary syphilis (Infections and infestations) | 7 (7) | 10 (11) | 0 (0)
Folliculitis (Infections and infestations) | 8 (16) | 8 (9) | 0 (0)
Conjunctivitis (Infections and infestations) | 6 (6) | 9 (10) | 0 (0)
Oral herpes (Infections and infestations) | 9 (13) | 6 (7) | 0 (0)
Gingivitis (Infections and infestations) | 9 (13) | 4 (4) | 0 (0)
Herpes zoster (Infections and infestations) | 8 (8) | 5 (5) | 0 (0)
Urethritis (Infections and infestations) | 8 (9) | 5 (5) | 0 (0)
Viral infection (Infections and infestations) | 4 (4) | 8 (8) | 0 (0)
Urethritis gonococcal (Infections and infestations) | 3 (4) | 8 (9) | 0 (0)
Cellulitis (Infections and infestations) | 8 (10) | 2 (3) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 (9) | 9 (10) | 0 (0)
Gastritis (Gastrointestinal disorders) | 9 (10) | 7 (7) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 5 (6) | 9 (13) | 0 (0)
Proctitis (Gastrointestinal disorders) | 6 (8) | 8 (9) | 0 (0)
Anogenital dysplasia (Gastrointestinal disorders) | 8 (10) | 4 (4) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 2 (5) | 9 (10) | 0 (0)
Dental caries (Gastrointestinal disorders) | 8 (8) | 2 (2) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 8 (10) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 6 (11) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (9) | 7 (12) | 0 (0)
Asthenia (General disorders) | 10 (12) | 14 (14) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 9 (10) | 6 (6) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 8 (8) | 3 (3) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 8 (8) | 3 (3) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 10 (11) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 8 (12) | 13 (15) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (9) | 11 (12) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (13) | 15 (17) | 0 (0)
Weight increased (Investigations) | 10 (10) | 9 (10) | 0 (0)
Hypertension (Vascular disorders) | 14 (16) | 5 (5) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 8 (8) | 6 (6) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 9 (9) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-06-14): https://cdn.clinicaltrials.gov/large-docs/64/NCT02831764/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-18): https://cdn.clinicaltrials.gov/large-docs/64/NCT02831764/SAP_002.pdf